CLINICAL TRIAL: NCT05052697
Title: A PHASE 1/2 RANDOMIZED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MODIFIED RNA VACCINE AGAINST INFLUENZA IN HEALTHY INDIVIDUALS
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Modified RNA Vaccine Against Influenza
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4781001
Record Dates: First submitted 2021-06-28; First posted 2021-09-22 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Influenza, Human
Keywords: Grippe; Flu; Influenza; Vaccine; RNA vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: SSA: observer-blinded, sponsor unblind SSB: single-blind, sponsor unblind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (28):
- SSA: mIRV A (dose level 1) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV A (dose level 2) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV A (dose level 3) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV A (dose level 4) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV B (dose level 1) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV B (dose level 2) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV B (dose level 3) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: mIRV B (dose level 4) + QIV (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: bIRV AB (dose level combination 1) + QIV (Experimental)
  Interventions: Biological: bIRV AB; Biological: QIV
- SSA: bIRV AB (dose level combination 2) + QIV (Experimental)
  Interventions: Biological: bIRV AB; Biological: QIV
- SSA: bIRV AB (dose level combination 3) + QIV (Experimental)
  Interventions: Biological: bIRV AB; Biological: QIV
- SSA: bIRV AB (dose level combination 4) + QIV (Experimental)
  Interventions: Biological: bIRV AB; Biological: QIV
- SSA: QIV + mIRV A strain (dose level 4) (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSA: qIRV (dose level 1) + QIV (Experimental)
  Interventions: Biological: qIRV; Biological: QIV
- SSA: QIV + mIRV B strain (dose level 4) (Experimental)
  Interventions: Biological: mIRV; Biological: QIV
- SSB: 2 doses of qIRV (dose level 1), 2-visit schedule (Experimental)
  Interventions: Biological: qIRV
- SSB: 2 doses of QIV, 2-visit schedule (Experimental)
  Interventions: Biological: QIV
- SSB: QIV + bIRV AA (dose level combination 1), 2-visit schedule (Experimental)
  Interventions: Biological: QIV; Biological: bIRV AA
- SSB: QIV + bIRV AA (dose level combination 2), 2-visit schedule (Experimental)
  Interventions: Biological: QIV; Biological: bIRV AA
- SSB: QIV + bIRV AA (dose level combination 1), 1-visit schedule (Experimental)
  Interventions: Biological: QIV; Biological: bIRV AA
- SSB: QIV + bIRV AA (dose level combination 2), 1-visit schedule (Experimental)
  Interventions: Biological: QIV; Biological: bIRV AA
- SSB: qIRV (dose level 2, dose combination 1), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered.
  Interventions: Biological: qIRV
- SSB: qIRV (dose level 2, dose combination 2), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered
  Interventions: Biological: qIRV
- SSB: qIRV (dose level 3), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered
  Interventions: Biological: qIRV
- SSB: bIRV AA + bIRV BB (both dose level combination 1), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered
  Interventions: Biological: bIRV AA; Biological: bIRV BB
- SSB: 1 dose of QIV, 1-visit schedule (Experimental): NOTE: Arm Description has not been entered
  Interventions: Biological: QIV
- SSB: qIRV (dose level 1), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered.
  Interventions: Biological: qIRV
- SSB: qIRV (dose level 2), 1-visit schedule (Experimental): NOTE: Arm Description has not been entered.
  Interventions: Biological: qIRV

INTERVENTIONS:
Biological: mIRV — Intramuscular injection
  Arms: SSA: QIV + mIRV A strain (dose level 4); SSA: QIV + mIRV B strain (dose level 4); SSA: mIRV A (dose level 1) + QIV; SSA: mIRV A (dose level 2) + QIV; SSA: mIRV A (dose level 3) + QIV; SSA: mIRV A (dose level 4) + QIV; SSA: mIRV B (dose level 1) + QIV; SSA: mIRV B (dose level 2) + QIV; SSA: mIRV B (dose level 3) + QIV; SSA: mIRV B (dose level 4) + QIV
Biological: bIRV AB — Intramuscular injection
  Arms: SSA: bIRV AB (dose level combination 1) + QIV; SSA: bIRV AB (dose level combination 2) + QIV; SSA: bIRV AB (dose level combination 3) + QIV; SSA: bIRV AB (dose level combination 4) + QIV
Biological: qIRV — Intramuscular injection
  Arms: SSA: qIRV (dose level 1) + QIV; SSB: 2 doses of qIRV (dose level 1), 2-visit schedule; SSB: qIRV (dose level 1), 1-visit schedule; SSB: qIRV (dose level 2), 1-visit schedule; SSB: qIRV (dose level 2, dose combination 1), 1-visit schedule; SSB: qIRV (dose level 2, dose combination 2), 1-visit schedule; SSB: qIRV (dose level 3), 1-visit schedule
Biological: QIV — Intramuscular injection
  Arms: SSA: QIV + mIRV A strain (dose level 4); SSA: QIV + mIRV B strain (dose level 4); SSA: bIRV AB (dose level combination 1) + QIV; SSA: bIRV AB (dose level combination 2) + QIV; SSA: bIRV AB (dose level combination 3) + QIV; SSA: bIRV AB (dose level combination 4) + QIV; SSA: mIRV A (dose level 1) + QIV; SSA: mIRV A (dose level 2) + QIV; SSA: mIRV A (dose level 3) + QIV; SSA: mIRV A (dose level 4) + QIV; SSA: mIRV B (dose level 1) + QIV; SSA: mIRV B (dose level 2) + QIV; SSA: mIRV B (dose level 3) + QIV; SSA: mIRV B (dose level 4) + QIV; SSA: qIRV (dose level 1) + QIV; SSB: 1 dose of QIV, 1-visit schedule; SSB: 2 doses of QIV, 2-visit schedule; SSB: QIV + bIRV AA (dose level combination 1), 1-visit schedule; SSB: QIV + bIRV AA (dose level combination 1), 2-visit schedule; SSB: QIV + bIRV AA (dose level combination 2), 1-visit schedule; SSB: QIV + bIRV AA (dose level combination 2), 2-visit schedule
Biological: bIRV AA — Intramuscular injection
  Arms: SSB: QIV + bIRV AA (dose level combination 1), 1-visit schedule; SSB: QIV + bIRV AA (dose level combination 1), 2-visit schedule; SSB: QIV + bIRV AA (dose level combination 2), 1-visit schedule; SSB: QIV + bIRV AA (dose level combination 2), 2-visit schedule; SSB: bIRV AA + bIRV BB (both dose level combination 1), 1-visit schedule
Biological: bIRV BB — Intramuscular injection
  Arms: SSB: bIRV AA + bIRV BB (both dose level combination 1), 1-visit schedule

SUMMARY:
This study will be divided into two substudies - Substudy A (SSA) and Substudy B (SSB)

Substudy A This is a Phase 1 randomized substudy to evaluate the safety and immunogenicity of monovalent influenza modRNA vaccine (mIRV) and bivalent influenza modRNA vaccine (bIRV) at various dose levels, and quadrivalent influenza modRNA vaccine (qIRV), in participants 65 to 85 years of age. Participants will receive at Vaccination 1 either:

* 1 of 4 dose levels of mIRV (either A or B Strain),
* 1 of 4 dose levels of bIRV (containing both A and B strains),
* qIRV (at 1 dose level), or
* A licensed quadrivalent influenza vaccine (QIV).

At approximately 8 weeks following Vaccination 1, participants will be unblinded and QIV (Vaccination 2) administered to participants not having previously received this at Vaccination 1. Additionally, participants who previously received QIV at Vaccination 1 will receive one of the following for Vaccination 2:

* mIRV encoding A strain at dose level 4, or
* mIRV encoding B strain at dose level 4.

Substudy B

This is a randomized substudy to evaluate the safety and immunogenicity of the following vaccination schedules in participants 65 to 85 years of age:

2-Visit Schedules

* 2 doses of qIRV (at a dose level 1), administered 21 days apart.
* 2 doses of licensed QIV, administered 21 days apart (as a control group)
* A dose of licensed QIV following by a dose of bIRV encoding 2 A strains at dose level combination 1 or 2, administered 21 days apart.

  1-Visit Schedules
* A dose of licensed QIV administered concurrently in the opposite arm with bIRV encoding 2 A strains at dose level combination 1 or 2.
* A dose of bIRV encoding 2 A strains administered concurrently in the opposite arm with a dose of bIRV encoding 2 B strains.at dose level 1.
* A dose of qIRV encoding 2 A strains and 2 B strains at dose level 2 (at one of two possible dose level combinations).
* A dose of qIRV encoding 2 A strains and 2 B strains at dose level 3.
* 1 dose of licensed QIV (as a control group).

Substudy B

In participants 18 to 64 years of age:

-A dose of qIRV encoding 2 A strains and 2 B strains at a dose level combination 1 or 2.

ELIGIBILITY:
Substudy A

Inclusion Criteria:

* Male or female participants 65 to 85 years of age.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Male participant who is able to father children and willing to use an acceptable method of contraception; or female participant not of childbearing potential; or male participant not able to father children.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Allergy to egg proteins (egg or egg products) or chicken proteins.
* Participant who has had significant exposure to laboratory-confirmed SARS-CoV-2 infection, COVID-19, or influenza in the past 14 days known prior to Visit 1
* Any participant who has a SARS-CoV-2 RT-PCR or antigen test in the past 10 days prior to Visit 1 that has not been confirmed as negative.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
* Vaccination with any influenza vaccine within 6 months (175 days) before study intervention administration.
* Any participant who has received or plans to receive a modRNA-platform SARS-CoV-2 vaccine within 60 days of Visit 1
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Screening hematology/blood chemistry lab >=Grade 1 abnormality. Except Bilirubin, other stable Grade1 abnormalities may be considered eligible by Investigator.
* Screening ECG that is consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or study results.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participation in strenuous or endurance exercise through Visit 3.
* Prior history of heart disease.

Substudy B

Inclusion Criteria:

* Male or female participants 65 to 85 years of age or .Male or female participants 18 to 64 years of age
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* For participants 65 to 85 years of age at the time of enrollment, receipt of licensed influenza vaccination for the 2021-2022 northern hemisphere season >4 months (120 days) before study intervention administration.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Allergy to egg proteins (egg or egg products) or chicken proteins.
* Participant who has had significant exposure to laboratory-confirmed SARS-CoV-2 infection, COVID-19, or influenza in the past 14 days known prior to Visit 201
* Any participant who has a SARS-CoV-2 RT-PCR or antigen test in the past 10 days prior to Visit 201 that has not been confirmed as negative.
* Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
* Any participant who has received or plans to receive a modRNA-platform SARS-CoV-2 vaccine within 28 days of Visit 201
* Any participant who has received licensed influenza vaccination for the 2022-2023 northern hemisphere influenza season.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
* Participation in strenuous or endurance exercise through Visit 205.
* Prior history of heart disease.
* Any abnormal screening troponin I laboratory value
* Screening 12-lead ECG that, as judged by the investigator, is consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1158 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (98):
- United States (98):
  - North Alabama Research Center, Athens, Alabama
  - The Heart Center, Athens, Alabama
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - Inland Valley Cardiovascular Center, Murrieta, California
  - Orange County Heart Institute, Orange, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Orange County Research Center, Tustin, California
  - Pediatrics-Infectious Diseases - Clinical Trials Center at University of Colorado Anschutz Medical C, Aurora, Colorado
  - UCHealth Heart and Vascular Center - Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale Cardiology, New Haven, Connecticut
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Halifax Health Medical Center, Daytona Beach, Florida
  - NYU Langone Cardiology Associates, Delray Beach, Florida
  - First Coast Heart & Vascular Center, Fleming Island, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Alliance for Multispecialty Research, LLC, Fort Myers, Florida
  - Millennium Physician Group, Fort Myers, Florida
  - Robert B. Pritt, DO, Fort Myers, Florida
  - Direct Helpers Research Center., Hialeah, Florida
  - Best Quality Research,Inc., Hialeah, Florida
  - Elixia Infectious Disease, LLC, Hollywood, Florida
  - First Coast Heart & Vascular Center, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Premier Cardiology and Vascular Associates, Maitland, Florida
  - LMG Research, Miami, Florida
  - Millennium Clinical Research, Miami, Florida
  - Optimus U Corporation, Miami, Florida
  - Suncoast Research Group, Miami, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Dr Gerardo A. Polanco, MD, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Jackson Medical Group Cardiac Care, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Central Florida Cardiology Group, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - My Cardiologist, South Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - IACT Health, Columbus, Georgia
  - IACT Health, Rincon, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - University of Iowa, Iowa City, Iowa
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Heartland Cardiology, LLC, Wichita, Kansas
  - Centennial Medical Group, Elkridge, Maryland
  - Associates of Cardiology, Silver Spring, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Pioneer Heart Institute, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Meridian Clinical Research - 3345 North 107th Street, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Sanjay Vohra, MD, F.A.C.C., Henderson, Nevada
  - Wr-Crcn, Llc., Las Vegas, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Penn Medicine, Somers Point, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - NYU Langone - Center for the Prevention of Cardiovascular Disease, New York, New York
  - NYU Langone Health, New York, New York
  - Rochester General Hospital Infectious Disease, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Upstate Health Care Center-University Cardiovascular Group of Syracuse, Syracuse, New York
  - SUNY Upstate Medical University Global Health Research Unit, Syracuse, New York
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Columbus Cardiovascular Associates, Inc, Columbus, Ohio
  - Pennsylvania Heart and Vascular Group, Jenkintown, Pennsylvania
  - Main Street Physician's Care, Little River, South Carolina
  - Prolato Clinical Research Center, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - DM Clinical Research, Humble, Texas
  - Cedar Health Research, Irving, Texas
  - Harmony Heart Group, Plano, Texas
  - Mt Olympus Medical Research, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Northwest Heart Center, Tomball, Texas
  - Centricity Research Suffolk Primary Care, Suffolk, Virginia
  - Sentara BelleHarbour, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Branche A, Mulligan MJ, Maniar A, Puente O, Oladipupo I, Crowther G, Zareba AM, Yi Z, Scully I, Gomme E, Koury K, Kitchin N, Allen PS, Anderson AS, Gurtman A, Lindert K. A Phase 1/2 Randomized Study to Evaluate the Safety, Tolerability, and Immunogenicity of Nucleoside-Modified Messenger RNA Influenza Vaccines in Healthy Adults. Vaccines (Basel). 2025 Apr 3;13(4):383. doi: 10.3390/vaccines13040383. PMID 40333267
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4781001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 2 substudies-Substudy A and Substudy B.
Pre-assignment Details: A total of 1158 participants (substudy A: 256+ substudy B: 902) were enrolled and randomized to receive study treatment.
Groups:
- SSA: mIRV A (Dose Level 1) + QIV: Participants received a single injection of monovalent influenza modified ribonucleic acid, (modRNA) vaccine (mIRV) encoding A strain at dose level 1, intramuscularly into the deltoid muscle at Day 1 (vaccination 1). Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV A (Dose Level 2) + QIV: Participants received a single injection of mIRV encoding A strain at dose level 2, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV A (Dose Level 3) + QIV: Participants received a single injection of mIRV encoding A strain at dose level 3, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV A (Dose Level 4) + QIV: Participants received a single injection of mIRV encoding A strain at dose level 4, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV A - Licensed QIV: Participants received a single injection of quadrivalent influenza vaccine (QIV), licensed, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of either mIRV A or B at dose level 4 (vaccination 2).
- SSA: mIRV B (Dose Level 1) + QIV: Participants received a single injection of mIRV encoding B strain at dose level 1, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV B (Dose Level 2) + QIV: Participants received a single injection of mIRV encoding B strain at dose level 2, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV B (Dose Level 3) + QIV: Participants received a single injection of mIRV encoding B strain at dose level 3, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV B (Dose Level 4) + QIV: Participants received a single injection of mIRV encoding B strain at dose level 4, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: mIRV B - Licensed QIV: Participants received a single injection of QIV, licensed, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose injection of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
- SSA: bIRV AB (Dose Level Combination 1) + QIV: Participants received a single injection of bivalent influenza modified RNA vaccine (bIRV) encoding A and B strains at dose level combination 1, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: bIRV AB (Dose Level Combination 2) + QIV: Participants received a single injection of bIRV encoding A and B strains at dose level combination 2, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: bIRV AB (Dose Level Combination 3) + QIV: Participants received a single injection of bIRV encoding A and B strains at dose level combination 3, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: bIRV AB (Dose Level Combination 4) + QIV: Participants received a single injection of bIRV encoding A and B strains at dose level combination 4, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: bIRV AB-Licensed QIV: Participants received a single injection of licensed quadrivalent influenza vaccine (QIV), intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular injection of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
- SSA: qIRV (Dose Level 1) + QIV: Participants received a single injection of quadrivalent influenza mod RNA vaccine (qIRV) - encoding 2A strains and 2B strains at a dose level 1 per strain, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of licensed QIV (vaccination 2).
- SSA: qIRV - Licensed QIV: Participants received a single injection of licensed QIV, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, the licensed QIV control group received either a single intramuscular dose of injection of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
- SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received intramuscular injections with 2 doses qIRV at dose level 1 administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding AA strains at dose level combination 1 administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding AA strains at dose level combination 2 administered 21 days apart as a part of initial enrollment.
- SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received two doses of licensed QIV administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as part of initial enrollment.
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 2) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, dose combination 2 administered at day 1 as a part of initial enrollment.
- SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of bIRV AA + bIRV BB both dose level combination 1 administered at day 1 as a part of initial enrollment.
- SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV as part of initial enrollment.
- SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 3 administered at day 1 as a part of initial enrollment.
- SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment: Participants aged 18 to 64 years received a single intramuscular injection of qIRV dose level 1 as a part of expanded enrollment.
- SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment: Participants aged 18 to 64 years received a single intramuscular injection of qIRV dose level 2 as a part of expanded enrollment.
- SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 1 as a part of expanded enrollment
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) at Day 1 as part of expanded enrollment.
- SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV as a part of expanded enrollment.
- SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment: Participants aged 65 to 85 years received intramuscular injections with 2 doses qIRV at dose Level 1 administered 21 days apart as a part of expanded enrollment.
Period: Substudy A
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Started | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination 1 | 15 | 15 | 15 | 14 | 15 | 15 | 15 | 16 | 14 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination 2 | 6 | 10 | 9 | 12 | 1 | 6 | 7 | 6 | 2 | 1 | 6 | 11 | 6 | 9 | 6 | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Indicates participants randomized to either mIRV A, mIRV B, bIRV A, bIRV B or qIRV and received licensed QIV at vaccination 2. Also, includes participants who were randomized to 'Licensed QIV' and received either 'mIRV A or mIRV B at dose level 4' at vaccination 2.) | 15 | 15 | 15 | 14 | 15 | 14 | 15 | 16 | 14 | 15 | 15 | 15 | 15 | 14 | 15 | 13 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not vaccinated | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SubStudy B: Initial Enrollment
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Started (Participants who were randomized) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 15 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 14 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination 2 (Included participants who were randomized to 2-Visit vaccination schedule) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 15 | 16 | 1 (Participant received vaccination 2 in error) | 0 (Participants not applicable to receive the vaccination) | 0 (Participants not applicable to receive the vaccination) | 0 (Participants not applicable to receive the vaccination) | 0 (Participants not applicable to receive the vaccination) | 0 (Participants not applicable to receive the vaccination) | 0 (Participants not applicable to receive the vaccination) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 14 | 14 | 16 | 15 | 13 | 16 | 16 | 14 | 15 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not vaccinated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy B: Expanded Enrollment
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Started (Participants who were randomized) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 132 | 133 | 117 | 117 | 115 | 117
Vaccination 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 131 | 131 | 116 | 117 | 115 | 117
Vaccination 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 101
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 128 | 130 | 110 | 111 | 109 | 117
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 7 | 6 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 2 | 0
Not completed — Refused study procedure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Not vaccinated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: SSA=Vaccination 1 safety population(pop):participants (par) who received vaccination 1. SSB=safety pop:par who received study intervention. Par were analyzed according to vaccine administered.1 par randomized to mIRV A(dose level3)+QIV received mIRV A(dose level1)+QIV.1 par randomized to mIRV B (dose level2)+QIV and mIRV B(dose level 3)+QIV received mIRV B(dose level 1)+QIV each.1 par randomized to bIRV AB(dose level combination 1)+QIV received bIRV AB(dose level combination 2)+QIV.
Groups:
- Total: Total of all reporting groups
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment | Total
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15 | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 14 | 15 | 15 | 131 | 131 | 116 | 117 | 115 | 117 | 1149
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=18 years | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15 | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 14 | 15 | 15 | 131 | 131 | 116 | 117 | 115 | 117 | 1149
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 4 | 6 | 7 | 11 | 10 | 9 | 11 | 7 | 7 | 12 | 6 | 7 | 10 | 8 | 10 | 8 | 8 | 6 | 9 | 8 | 8 | 7 | 8 | 7 | 9 | 77 | 74 | 61 | 60 | 67 | 65 | 629
  Male | 8 | 8 | 7 | 10 | 9 | 10 | 3 | 5 | 5 | 4 | 7 | 9 | 3 | 9 | 8 | 5 | 7 | 4 | 7 | 8 | 10 | 7 | 7 | 8 | 9 | 6 | 8 | 6 | 54 | 57 | 55 | 57 | 48 | 52 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 2 | 7 | 3 | 5 | 5 | 3 | 8 | 5 | 4 | 4 | 4 | 4 | 4 | 12 | 9 | 9 | 10 | 8 | 8 | 12 | 10 | 11 | 9 | 14 | 74 | 77 | 50 | 60 | 55 | 55 | 546
  Not Hispanic or Latino | 13 | 14 | 13 | 13 | 13 | 10 | 11 | 10 | 9 | 11 | 6 | 11 | 11 | 11 | 11 | 11 | 10 | 2 | 6 | 7 | 6 | 8 | 7 | 4 | 6 | 3 | 6 | 1 | 57 | 54 | 65 | 56 | 60 | 62 | 598
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 1 | 1 | 2 | 1 | 1 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Black or African American | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 4 | 2 | 4 | 3 | 1 | 2 | 4 | 1 | 2 | 1 | 20 | 20 | 21 | 12 | 14 | 11 | 143
  White | 14 | 14 | 14 | 13 | 13 | 13 | 13 | 12 | 14 | 14 | 13 | 15 | 14 | 15 | 12 | 13 | 13 | 13 | 10 | 14 | 11 | 12 | 13 | 14 | 12 | 13 | 11 | 14 | 98 | 107 | 92 | 101 | 96 | 104 | 964
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 3 | 0 | 8
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination 1: Substudy A
Description: Local reactions included pain at the injection site, redness and swelling and were recorded by participants in an electronic diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as mild (Grade 1): greater than (>) 2.0 cm to 5.0 cm; moderate (Grade 2): >5.0 cm to 10.0 cm; severe (Grade 3): >10 cm; potentially life-threatening (Grade 4): necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild (Grade 1): did not interfere with activity; moderate (Grade 2): interfered with activity; severe (Grade 3): prevented daily activity and potentially life-threatening (Grade 4): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Exact 2-sided confidence interval was based on the Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after Vaccination 1
Population: Vaccination 1 safety population included all the participants who received vaccination 1. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 14 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Redness: Mild | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 14.3 [1.8 to 42.8] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9]
  Redness: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Redness: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Redness: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Swelling: Mild | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9]
  Swelling: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Swelling: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Swelling: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Pain at injection site: Mild | 25.0 [7.3 to 52.4] | 33.3 [11.8 to 61.6] | 42.9 [17.7 to 71.1] | 50.0 [23.0 to 77.0] | 53.3 [26.6 to 78.7] | 29.4 [10.3 to 56.0] | 28.6 [8.4 to 58.1] | 42.9 [17.7 to 71.1] | 28.6 [8.4 to 58.1] | 40.0 [16.3 to 67.7] | 42.9 [17.7 to 71.1] | 25.0 [7.3 to 52.4] | 53.3 [26.6 to 78.7] | 46.7 [21.3 to 73.4] | 40.0 [16.3 to 67.7] | 80.0 [51.9 to 95.7] | 53.3 [26.6 to 78.7]
  Pain at injection site: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5]
  Pain at injection site: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Pain at injection site: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]

2. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination 2: Substudy A
Description: Local reactions included pain at the injection site, redness and swelling and were recorded by participants in an electronic diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 cm. Redness and swelling were graded as mild (Grade 1): >2.0 cm to 5.0 cm; moderate (Grade 2): >5.0 cm to 10.0 cm; severe (Grade 3): >10 cm; potentially life-threatening (Grade 4): necrosis or exfoliative dermatitis. Pain at injection site was graded as mild (Grade 1): did not interfere with activity; moderate (Grade 2): interfered with activity; severe (Grade 3): prevented daily activity and potentially life-threatening (Grade 4): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Exact 2-sided confidence interval was based on the Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after Vaccination 2
Population: Vaccination 2 safety population included all the participants who received vaccination 2. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure. Data for mIRV A + Licensed QIV is missing as there was no e-diary data transmitted.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Licensed QIV + mIRV A Strain (Dose Level 4): Participants who received Licensed QIV as Vaccination 1, were administered mIRV A- dose level 4, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- Licensed QIV + mIRV B Strain (Dose Level 4): Participants who received Licensed QIV, as Vaccination 1, were administered mIRV B at dose level 4, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- mIRV A + Licensed QIV: Participants who received mIRV-A as Vaccination 1, were administered Licensed QIV, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- mIRV B + Licensed QIV: Participants who received mIRV B as Vaccination 1, were administered Licensed QIV intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- bIRV AB + Licensed QIV: Participants who received bIRV AB as Vaccination 1, were administered Licensed QIV, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- qIRV + Licensed QIV: Participants who received qIRV as Vaccination 1, were administered Licensed QIV intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
Arm/Group | Licensed QIV + mIRV A Strain (Dose Level 4) | Licensed QIV + mIRV B Strain (Dose Level 4) | mIRV A + Licensed QIV | mIRV B + Licensed QIV | bIRV AB + Licensed QIV | qIRV + Licensed QIV
Number analyzed (Participants) | 8 | 3 | 0 | 7 | 23 | 6
Percentage of participants
  Redness: Mild | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 14.3 [0.4 to 57.9] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  Redness: Moderate | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] |  | 0 [0.0 to 41.0] | 8.7 [1.1 to 28.0] | 0 [0.0 to 45.9]
  Redness: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Redness: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Swelling: Mild | 12.5 [0.3 to 52.7] | 0 [0.0 to 70.8] |  | 14.3 [0.4 to 57.9] | 0 [0.0 to 14.8] | 16.7 [0.4 to 64.1]
  Swelling: Moderate | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  Swelling: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Swelling: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Pain at injection site: Mild | 50.0 [15.7 to 84.3] | 33.3 [0.8 to 90.6] |  | 57.1 [18.4 to 90.1] | 30.4 [13.2 to 52.9] | 50.0 [11.8 to 88.2]
  Pain at injection site: Moderate | 12.5 [0.3 to 52.7] | 66.7 [9.4 to 99.2] |  | 14.3 [0.4 to 57.9] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Pain at injection site: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  Pain at injection site: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]

3. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination 1: Substudy A
Description: Systemic events included fever, vomiting, diarrhea, headache,fatigue,chills,new/worsened muscle pain & new/worsened joint pain & recorded by participants in an electronic diary.Fever defined as oral temperature greater than equal to(>=)38.0 degrees Celsius(deg C) & categorized as>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C,>38.9 to 40.0 deg C & >40.0 deg C. Vomiting graded as:Grade(G)1:1-2 times in 24 hours(h);G2:>2 times in 24h;G3:required Intravenous (IV) hydration.Diarrhea graded as: G1:2-3 loose stools in 24h;G2: 4-5 loose stools in 24h;G3: 6 or more loose stools in 24h.Headache,fatigue,chills, new/worsened muscle pain & new/worsened joint pain:G1:didn't interfere with activity;G2: some interference with activity;G3:prevented daily routine activity.For all systemic events except fever, Grade 4=emergency room visit or hospitalization. Grade 4 events were classified by the investigator or medically qualified person.Exact 2-sided confidence interval based on Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 After Vaccination 1
Population: Vaccination 1 safety population included all participants who received the study vaccination 1. 'Number Analyzed' signifies number of participants evaluable for the specified rows. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 14 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Fever: >=38.0 deg C to 38.4 deg C | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Fever: >38.4 deg C to 38.9 deg C | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Fever: >40.0 deg C | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Fatigue: Mild | 18.8 [4.0 to 45.6] | 0 [0.0 to 21.8] | 14.3 [1.8 to 42.8] | 35.7 [12.8 to 64.9] | 6.7 [0.2 to 31.9] | 11.8 [1.5 to 36.4] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 21.4 [4.7 to 50.8] | 13.3 [1.7 to 40.5] | 28.6 [8.4 to 58.1] | 18.8 [4.0 to 45.6] | 13.3 [1.7 to 40.5] | 46.7 [21.3 to 73.4] | 13.3 [1.7 to 40.5] | 26.7 [7.8 to 55.1] | 33.3 [11.8 to 61.6]
  Fatigue: Moderate | 12.5 [1.6 to 38.3] | 13.3 [1.7 to 40.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 14.3 [1.8 to 42.8] | 14.3 [1.8 to 42.8] | 14.3 [1.8 to 42.8] | 26.7 [7.8 to 55.1] | 7.1 [0.2 to 33.9] | 6.3 [0.2 to 30.2] | 26.7 [7.8 to 55.1] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5] | 13.3 [1.7 to 40.5] | 20.0 [4.3 to 48.1]
  Fatigue: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Fatigue: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Headache: Mild | 12.5 [1.6 to 38.3] | 13.3 [1.7 to 40.5] | 7.1 [0.2 to 33.9] | 21.4 [4.7 to 50.8] | 6.7 [0.2 to 31.9] | 5.9 [0.1 to 28.7] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 7.1 [0.2 to 33.9] | 33.3 [11.8 to 61.6] | 14.3 [1.8 to 42.8] | 6.3 [0.2 to 30.2] | 20.0 [4.3 to 48.1] | 6.7 [0.2 to 31.9] | 20.0 [4.3 to 48.1] | 26.7 [7.8 to 55.1] | 13.3 [1.7 to 40.5]
  Headache: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 11.8 [1.5 to 36.4] | 21.4 [4.7 to 50.8] | 0 [0.0 to 23.2] | 14.3 [1.8 to 42.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8]
  Headache: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Headache: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Chills: Mild | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 26.7 [7.8 to 55.1] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 6.7 [0.2 to 31.9]
  Chills: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Chills: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Chills: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Vomiting: Mild | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Vomiting: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Vomiting: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Vomiting: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Diarrhea: Mild | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 14.3 [1.8 to 42.8] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 20.6] | 20.0 [4.3 to 48.1] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5]
  Diarrhea: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Diarrhea: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  Diarrhea: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  New or worsened muscle pain: Mild | 18.8 [4.0 to 45.6] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 12.5 [1.6 to 38.3] | 20.0 [4.3 to 48.1] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 21.8]
  New or worsened muscle pain: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 5.9 [0.1 to 28.7] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 6.3 [0.2 to 30.2] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5]
  New or worsened muscle pain: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  New or worsened joint pain: Mild | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 0 [0.0 to 23.2] | 13.3 [1.7 to 40.5] | 14.3 [1.8 to 42.8] | 6.3 [0.2 to 30.2] | 20.0 [4.3 to 48.1] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 21.8] | 6.7 [0.2 to 31.9]
  New or worsened joint pain: Moderate | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8]
  New or worsened joint pain: Severe | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 19.5] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8]

4. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination 2: Substudy A
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, chills, new/worsened muscle pain & new /worsened joint pain & recorded by participants in electronic diary. Fever defined as oral temperature >=38.0 deg C & categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C & >40.0 deg C. Vomiting graded as: Grade(G) 1: 1-2 times in 24 h; G2: >2 times in 24 h; G3: required IV hydration. Diarrhea graded as: G1: 2-3 loose stools in 24 h; G2: 4-5 loose stools in 24 h; G3: 6 or more loose stools in 24 h. Headache, fatigue, chills, new/worsened muscle pain & new/worsened joint pain: G1: didn't interfere with activity; G2: some interference with activity; G3: prevented daily routine activity. For all systemic events except fever, Grade 4= emergency room visit or hospitalization. Grade 4 events were classified by the investigator or medically qualified person. Exact 2-sided confidence interval based on Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after Vaccination 2
Population: Vaccination 2 safety population included all participants who received vaccination 2. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows. Data for mIRV A + Licensed QIV is missing as there was no e-diary data transmitted.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Licensed QIV + mIRV B Strain (Dose Level 4): Participants who received Licensed QIV, Vaccination 1, were administered mIRV- B at dose level 4, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
- mIRV B + Licensed QIV: Participants who received mIRV-B as Vaccination 1, were administered Licensed QIV, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
Arm/Group | Licensed QIV + mIRV A Strain (Dose Level 4) | Licensed QIV + mIRV B Strain (Dose Level 4) | mIRV A + Licensed QIV | mIRV B + Licensed QIV | bIRV AB + Licensed QIV | qIRV + Licensed QIV
Number analyzed (Participants) | 8 | 3 | 0 | 7 | 23 | 6
Percentage of participants
  Fever: >=38.0 deg C to 38.4 deg C | 12.5 [0.3 to 52.7] | 66.7 [9.4 to 99.2] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Fever: >38.4 deg C to 38.9 deg C | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Fever: >40.0 deg C | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Fatigue: Mild | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 42.9 [9.9 to 81.6] | 13.0 [2.8 to 33.6] | 0 [0.0 to 45.9]
  Fatigue: Moderate | 25.0 [3.2 to 65.1] | 100.0 [29.2 to 100.0] |  | 14.3 [0.4 to 57.9] | 8.7 [1.1 to 28.0] | 0 [0.0 to 45.9]
  Fatigue: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Fatigue: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Headache: Mild | 12.5 [0.3 to 52.7] | 33.3 [0.8 to 90.6] |  | 28.6 [3.7 to 71.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  Headache: Moderate | 12.5 [0.3 to 52.7] | 33.3 [0.8 to 90.6] |  | 0 [0.0 to 41.0] | 13.0 [2.8 to 33.6] | 0 [0.0 to 45.9]
  Headache: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Headache: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Chills: Mild | 12.5 [0.3 to 52.7] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Chills: Moderate | 0 [0.0 to 36.9] | 66.7 [9.4 to 99.2] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  Chills: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Chills: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Vomiting: Mild | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Vomiting: Moderate | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Vomiting: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Vomiting: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Diarrhea: Mild | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 14.3 [0.4 to 57.9] | 0 [0.0 to 14.8] | 16.7 [0.4 to 64.1]
  Diarrhea: Moderate | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Diarrhea: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  Diarrhea: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Mild | 12.5 [0.3 to 52.7] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Moderate | 0 [0.0 to 36.9] | 33.3 [0.8 to 90.6] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  New or worsened joint pain: Mild | 0 [0.0 to 36.9] | 0.0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  New or worsened joint pain: Moderate | 12.5 [0.3 to 52.7] | 66.7 [9.4 to 99.2] |  | 0 [0.0 to 41.0] | 4.3 [0.1 to 21.9] | 0 [0.0 to 45.9]
  New or worsened joint pain: Severe | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 36.9] | 0 [0.0 to 70.8] |  | 0 [0.0 to 41.0] | 0 [0.0 to 14.8] | 0 [0.0 to 45.9]

5. Primary Outcome: Percentage of Participants Reporting Adverse Events After Vaccination 1: Substudy A
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e, excluding local reactions and systematic events) were reported in this outcome measure.
Time Frame: From Day 1 up to 4 weeks After Vaccination 1
Population: Vaccination 1 safety population included all participants who received Vaccination 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants | 12.5 [1.6 to 38.3] | 20.0 [4.3 to 48.1] | 7.1 [0.2 to 33.9] | 14.3 [1.8 to 42.8] | 20.0 [4.3 to 48.1] | 17.6 [3.8 to 43.4] | 28.6 [8.4 to 58.1] | 13.3 [1.7 to 40.5] | 21.4 [4.7 to 50.8] | 6.7 [0.2 to 31.9] | 50.0 [23.0 to 77.0] | 18.8 [4.0 to 45.6] | 40.0 [16.3 to 67.7] | 13.3 [1.7 to 40.5] | 26.7 [7.8 to 55.1] | 20.0 [4.3 to 48.1] | 6.7 [0.2 to 31.9]

6. Primary Outcome: Percentage of Participants Reporting Adverse Events After Vaccination 2: Substudy A
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: From Day 1 up to 4 weeks After vaccination 2
Population: Vaccination 2 safety population included all participants who received Vaccination 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Licensed QIV + mIRV A Strain (Dose Level 4): Participants who received Licensed QIV, as Vaccination 1, were administered mIRV A at dose level 4, intramuscularly as Vaccination 2 at 8 weeks after Vaccination 1.
Arm/Group | Licensed QIV + mIRV A Strain (Dose Level 4) | Licensed QIV + mIRV B Strain (Dose Level 4) | mIRV A + Licensed QIV | mIRV B + Licensed QIV | bIRV AB + Licensed QIV | qIRV + Licensed QIV
Number analyzed (Participants) | 11 | 3 | 37 | 21 | 32 | 7
Percentage of participants | 9.1 [0.2 to 41.3] | 0 [0.0 to 70.8] | 8.1 [1.7 to 21.9] | 14.3 [3.0 to 36.3] | 25.0 [11.5 to 43.4] | 28.6 [3.7 to 71.0]

7. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAE) From First Vaccination to 6 Months After Last Vaccination: Substudy A
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event.
Time Frame: From vaccination 1 on day 1 up to 6 months after vaccination 2
Population: Safety population included all the participants who received the study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 5.9 | 0.0 | 0.0 | 0.0 | 6.7 | 7.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Percentage of Participants With Abnormal Hematology Values at 2 Days After Vaccination 1: Substudy A
Description: Hematology parameters included erythrocytes, lymphocytes, neutrophils, eosinophils/leukocytes, erythrocyte (ery) mean corpuscular volume, ery. mean corpuscular hemoglobin and ery. mean corpuscular hemoglobin concentration. The primary criteria were as follows erythrocytes, lymphocytes, neutrophils: <0.8*lower limit of normal (LLN); Lymphocytes/Leukocytes, Eosinophils/Leukocytes, Monocytes/Leukocytes: >1.2*upper limit of normal (ULN); Ery. Mean Corpuscular Volume:>1.1*ULN; Ery. Mean Corpuscular Hemoglobin and Ery.Mean Corpuscular hemoglobin Concentration: < 0.9*LLN. Also add 95% CI was based on Clopper and Pearson method.
Time Frame: 2 days after vaccination 1
Population: Vaccination 1 safety population included all participants who received vaccination 1. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Erythrocytes: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 13 | 15 | 15 | 14 | 15 | 14 | 15
  Erythrocytes | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8]
  Lymphocytes: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 13 | 15 | 15 | 14 | 15 | 14 | 15
  Lymphocytes | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9]
  Neutrophils: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 13 | 15 | 15 | 14 | 15 | 0 | 0
  Neutrophils | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] |  |
  Eosinophils/Leukocytes: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils/Leukocytes | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] |  |  |  |  |  |  |
  Monocytes/Leukocytes: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 13 | 15 | 15 | 14 | 15 | 14 | 15
  Monocytes/Leukocytes | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 7.7 [0.2 to 36.0] | 28.6 [8.4 to 58.1] | 0 [0.0 to 21.8] | 13.3 [1.7 to 40.5] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 24.7] | 6.7 [0.2 to 31.9] | 7.7 [0.2 to 36.0] | 13.3 [1.7 to 40.5] | 13.3 [1.7 to 40.5] | 14.3 [1.8 to 42.8] | 20.0 [4.3 to 48.1] | 14.3 [1.8 to 42.8] | 6.7 [0.2 to 31.9]
  Ery. Mean Corpuscular Volume: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Volume | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] |  |  |  |  |  |  |
  Ery. Mean Corpuscular Hemoglobin: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  Ery. Mean Corpuscular Hemoglobin | 6.7 [0.2 to 31.9] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] |  |  |  |  |  | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8]
  Ery. Mean Corpuscular HGB Concentration: number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 21.8] |  |  |  |  |  |  |

9. Primary Outcome: Percentage of Participants With Abnormal Hematology Values at 1 Week After Vaccination 1: Substudy A
Description: Hematology parameters included erythrocytes, neutrophils, eosinophils/leukocytes, monocytes/leukocytes, ery mean corpuscular hemoglobin. The primary criteria were as follows erythrocytes and neutrophils: <0.8* LLN; Eosinophils/Leukocytes and Monocytes/Leukocytes: >1.2* ULN; Ery. Mean Corpuscular Hemoglobin:>1.1*ULN. 95% CI was based on Clopper and Pearson method.
Time Frame: 1 week after vaccination 1
Population: Vaccination 1 safety population included all participants who received the study vaccination 1. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 14 | 14 | 15 | 14 | 16 | 15 | 15 | 14 | 15 | 14
Percentage of participants
  Erythrocytes: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Erythrocytes | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 7.7 [0.2 to 36.0] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 6.3 [0.2 to 30.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2]
  Neutrophils: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 16 | 15 | 15 | 14 | 0 | 0
  Neutrophils |  |  |  |  |  |  |  |  |  |  | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] |  |
  Eosinophils/Leukocytes: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Eosinophils/Leukocytes | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2]
  Monocytes/Leukocytes: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Monocytes/Leukocytes | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 20.6] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9]
  Ery. Mean Corpuscular Hemoglobin: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 0 | 0 | 0 | 0 | 0 | 15 | 14
  Ery. Mean Corpuscular Hemoglobin | 6.3 [0.2 to 30.2] | 0 [0.0 to 21.8] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 0 [0.0 to 20.6] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 0 [0.0 to 24.7] |  |  |  |  |  | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2]

10. Primary Outcome: Percentage of Participants With Abnormal Chemistry Values at 2 Days After Vaccination 1: Substudy A
Description: Chemistry parameters included blood urea nitrogen and C-reactive protein. The primary criteria were as follows Blood Urea Nitrogen: > 1.3*ULN; C Reactive Protein: > 1.1*ULN. 95% CI was based on Clopper and Pearson method.
Time Frame: 2 days after vaccination 1
Population: Vaccination 1 safety population included all participants who received vaccination 1. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 16 | 14 | 15 | 14 | 15 | 13 | 16 | 15 | 14 | 15 | 15 | 15
Percentage of participants
  Blood Urea Nitrogen | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 14.3 [1.8 to 42.8] | 6.7 [0.2 to 31.9] | 6.3 [0.2 to 30.2] | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 7.7 [0.2 to 36.0] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8]
  C Reactive Protein | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 14.3 [1.8 to 42.8] | 21.4 [4.7 to 50.8] | 26.7 [7.8 to 55.1] | 18.8 [4.0 to 45.6] | 7.1 [0.2 to 33.9] | 26.7 [7.8 to 55.1] | 30.8 [9.1 to 61.4] | 20.0 [4.3 to 48.1] | 15.4 [1.9 to 45.4] | 25.0 [7.3 to 52.4] | 40.0 [16.3 to 67.7] | 28.6 [8.4 to 58.1] | 20.0 [4.3 to 48.1] | 26.7 [7.8 to 55.1] | 20.0 [4.3 to 48.1]

11. Primary Outcome: Percentage of Participants With Abnormal Chemistry Values at 1 Week After Vaccination 1: Substudy A
Description: Chemistry parameters included blood urea nitrogen and C-reactive protein. The primary criteria were as follows Blood Urea Nitrogen: > 1.3*ULN; C Reactive Protein: > 1.1*ULN. Also add 95% CI was based on Clopper and Pearson method.
Time Frame: 1 week after vaccination 1
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 16 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Blood Urea Nitrogen | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 20.6] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 20.6] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 0 [0.0 to 21.8] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9]
  C-reactive protein: number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 14 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
  C-reactive protein | 0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 0 [0.0 to 23.2] | 0 [0.0 to 23.2] | 0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 6.7 [0.2 to 31.9] | 13.3 [1.7 to 40.5] | 0 [0.0 to 21.8]

12. Primary Outcome: Percentage of Participants With Grade Shifts in Hematology Values at 2 Days After Vaccination 1: Substudy A
Description: Hematology parameters included hemoglobin, lymphocytes, neutrophils decrease, platelets decrease, white blood cells (WBC) decrease and WBC increase. Laboratory abnormalities were graded by Food and Drug Administration (FDA) toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in hematology values were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 2 days after vaccination 1 were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported.
Time Frame: From Baseline (prior to vaccination 1) to 2 days after vaccination 1
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 15 | 15 | 13 | 14 | 15 | 15 | 14 | 14 | 13 | 15 | 13 | 15 | 15 | 14 | 15 | 14 | 15
Percentage of participants
  Hemoglobin: Baseline Normal to Grade 1 | 0 | 6.7 | 7.7 | 14.3 | 6.7 | 0 | 14.3 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 6.7 | 0 | 0
  Hemoglobin: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Baseline Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0
  Lymphocytes: Baseline Normal to Grade 1 | 0 | 6.7 | 15.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0
  Lymphocytes: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 1.7 | 0 | 0 | 0 | 0 | 0 | 6.7
  Neutrophil Decrease: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 6.7 | 0 | 0 | 0 | 7.1 | 0
  Platelets Decrease: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.7 | 0 | 0 | 0 | 0 | 0 | 0
  WBC decrease: Baseline Normal to Grade 1 | 0 | 6.7 | 7.7 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7
  WBC increase: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Percentage of Participants With Grade Shifts in Hematology Values at 1 Week After Vaccination 1: Substudy A
Description: Hematology parameters included hemoglobin, lymphocytes, neutrophils decrease, WBC decrease and WBC increase. Laboratory abnormalities were graded by FDA toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in hematology values were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 1 week after vaccination 1 were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported.
Time Frame: From Baseline (prior to vaccination 1) to 1 week after vaccination 1
Population: Vaccination 1 safety population included all participants who received vaccination 1. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 16 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  Hemoglobin: Baseline Normal to Grade 1: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Hemoglobin: Baseline Normal to Grade 1 | 0 | 0 | 7.7 | 7.1 | 0 | 6.3 | 14.3 | 0 | 0 | 0 | 7.1 | 6.3 | 0 | 6.7 | 0 | 0 | 0
  Hemoglobin: Baseline Normal to Grade 2: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Hemoglobin: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Baseline Normal to Grade 1: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Lymphocytes: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 7.7 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 6.7 | 7.1
  Lymphocytes: Baseline Grade 1 to Grade 2: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Lymphocytes: Baseline Grade 1 to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1
  Neutrophil decrease: Baseline Normal to Grade 1: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Neutrophil decrease: Baseline Normal to Grade 1 | 0 | 0 | 7.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil decrease: Baseline Normal to Grade 2: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Neutrophil decrease: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1
  Neutrophil decrease: Baseline Grade 2 to Grade 3: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  Neutrophil decrease: Baseline Grade 2 to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0
  WBC decrease: Baseline Normal to Grade 1: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  WBC decrease: Baseline Normal to Grade 1 | 0 | 0 | 7.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14.3
  WBC decrease: Baseline Normal to Grade 2: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  WBC decrease: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC increase: Baseline Normal to Grade 1: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  WBC increase: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC increase: Baseline Normal to Grade 2: number analyzed (Participants) | 16 | 15 | 13 | 14 | 15 | 16 | 14 | 13 | 14 | 13 | 14 | 16 | 15 | 15 | 14 | 15 | 14
  WBC increase: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Percentage of Participants With Grade Shifts in Chemistry Laboratory Values at 2 Days After Vaccination 1: Substudy A
Description: Chemistry abnormalities were graded by toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in chemistry values were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 2 days after vaccination 1 (post-baseline) were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported. The parameters reported were - Alanine Aminotransferase Increased (ALP), Alkaline Phosphatase Increased (ALP), Aspartate Aminotransferase Increased (AST), Creatinine Increased and Urea Nitrogen.
Time Frame: From Baseline (prior to vaccination 1) to 2 days after vaccination 1
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 16 | 14 | 15 | 14 | 15 | 13 | 16 | 15 | 14 | 15 | 15 | 15
Percentage of participants
  ALT Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7
  ALP Increased: Baseline Normal to Grade 1 | 0 | 1.67 | 0 | 0 | 0 | 0 | 14.3 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0
  AST Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14.3 | 0 | 0 | 6.3 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Baseline Normal to Grade 1 | 6.3 | 0 | 7.1 | 7.1 | 6.7 | 0 | 0 | 0 | 0 | 13.3 | 0 | 0 | 0 | 6.7 | 0 | 0 | 6.7
  Urea Nitrogen: Baseline Normal to Grade 2 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0
  Urea Nitrogen: Baseline Grade 1 to Grade 2 | 0 | 0 | 0 | 7.1 | 0 | 6.3 | 0 | 6.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Percentage of Participants With Grade Shifts in Chemistry Laboratory Values at 1 Week After Vaccination 1: Substudy A
Description: Chemistry abnormalities were graded by toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in chemistry values were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 1 week after vaccination 1 (post-baseline) were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported. The parameters reported were - Alanine Aminotransferase Increased, Alkaline Phosphatase Increased, Aspartate Aminotransferase Increased, Creatinine Increased and Urea Nitrogen.
Time Frame: From Baseline (prior to vaccination 1) to 1 week after vaccination 1
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 16 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants
  ALT Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 6.7
  ALP Increased: Baseline Normal to Grade 1 | 0 | 6.7 | 0 | 0 | 0 | 6.3 | 7.1 | 0 | 7.1 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 0
  AST Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13.3
  Creatinine Increased: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Baseline Normal to Grade 1 | 0 | 0 | 0 | 0 | 0 | 6.3 | 14.3 | 0 | 0 | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0
  Urea Nitrogen: Baseline Normal to Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Baseline Grade 1 to Grade 2 | 0 | 0 | 0 | 7.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Percentage of Participants With New Electrocardiogram (ECG) Abnormalities at 2 Days After Vaccination 1: Substudy A
Description: An ECG abnormality was defined as any new abnormality that, as judged by a cardiologist, was consistent with probable or possible myocarditis or pericarditis, including: Sustained atrial or ventricular arrhythmias, Second-degree Mobitz Type II or worse atrioventricular block, new bundle branch block and Diffuse ST-segment elevation or PR-segment inversion, compatible with pericarditis.
Time Frame: 2 days after vaccination 1
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

17. Primary Outcome: Percentage of Participants With New Electrocardiogram (ECG) Abnormalities at 1 Week After Vaccination 1: Substudy A
Description: as for outcome 16
Time Frame: 1 week after vaccination 1
Population: Vaccination 1 safety population included all participants who received vaccination 1.
Measure: Number; unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 16 | 15 | 14 | 14 | 15 | 17 | 14 | 15 | 14 | 15 | 14 | 16 | 15 | 15 | 15 | 15 | 15
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

18. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination for 1-Visit Schedule (Initial Enrollment): Substudy B
Description: Local reactions included pain at the injection site, redness and swelling and were recorded by participants in an electronic diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 cm. Redness and swelling were graded as mild (Grade 1): >2.0 cm to 5.0 cm; moderate (Grade 2): >5.0 cm to 10.0 cm; severe (Grade 3): >10 cm; potentially life-threatening (Grade 4): necrosis or exfoliative dermatitis. Pain at injection site was graded as mild (Grade 1): did not interfere with activity; moderate (Grade 2): interfered with activity; severe (Grade 3): prevented daily activity and potentially life-threatening (Grade 4): emergency room visit or hospitalization for severe pain. Exact 2-sided confidence interval was based on the Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Safety population included all the participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) at Day 1 as part of initial enrollment.
Arm/Group | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 14 | 16 | 15
Percentage of participants
  Redness: Mild | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 20.0 [4.3 to 48.1]
  Redness: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 14.3 [1.8 to 42.8] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9]
  Redness: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Redness: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Swelling: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9]
  Swelling: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8] | 14.3 [1.8 to 42.8] | 12.5 [1.6 to 38.3] | 0.0 [0.0 to 21.8]
  Swelling: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Swelling: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Pain at injection site: Mild | 31.3 [11.0 to 58.7] | 40.0 [16.3 to 67.7] | 31.3 [11.0 to 58.7] | 13.3 [1.7 to 40.5] | 14.3 [1.8 to 42.8] | 25.0 [7.3 to 52.4] | 33.3 [11.8 to 61.6]
  Pain at injection site: Moderate | 6.3 [0.2 to 30.2] | 20.0 [4.3 to 48.1] | 18.8 [4.0 to 45.6] | 0.0 [0.0 to 21.8] | 14.3 [1.8 to 42.8] | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9]
  Pain at injection site: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]

19. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination 1 for 2- Visit Schedule (Initial Enrollment): Substudy B
Description: as for outcome 18
Time Frame: From Day 1 to Day 7 after vaccination 1
Population: Safety population included all the participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16
Percentage of participants
  Redness: Mild | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 20.6]
  Redness: Moderate | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Redness: Severe | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Redness: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Swelling: Mild | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 20.6]
  Swelling: Moderate | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Swelling: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Swelling: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Pain at injection site: Mild | 21.4 [4.7 to 50.8] | 40.0 [16.3 to 67.7] | 31.3 [11.0 to 58.7] | 25.0 [7.3 to 52.4]
  Pain at injection site: Moderate | 28.6 [8.4 to 58.1] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Pain at injection site: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]

20. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination 2 for 2- Visit Schedule (Initial Enrollment): Substudy B
Description: as for outcome 18
Time Frame: From Day 1 to Day 7 after vaccination 2
Population: Safety population included all the participants who received the study intervention. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding 2A strains at dose level combination 2 administered 21 days apart as a part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 13 | 14 | 15 | 16
Percentage of participants
  Redness: Mild | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Redness: Moderate | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  Redness: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Redness: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Swelling: Mild | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Swelling: Moderate | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 6.3 [0.2 to 30.2]
  Swelling: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Swelling: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Pain at injection site: Mild | 30.8 [9.1 to 61.4] | 42.9 [17.7 to 71.1] | 13.3 [1.7 to 40.5] | 18.8 [4.0 to 45.6]
  Pain at injection site: Moderate | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  Pain at injection site: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]

21. Primary Outcome: Percentage of Participants Reporting Local Reactions After Vaccination for Expanded Enrollment: Substudy B
Description: as for outcome 18
Time Frame: From Day 1 to Day 7 after vaccination 1 for all arms; From Day 1 to Day 7 after vaccination 2 for 2 doses of qIRV (dose level 1), 2-visit schedule arm
Population: Safety population included all the participants who received the study intervention. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed'(n) = number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Participants aged 18 to 64 years received a single intramuscular injection of qIRV dose level 2 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 131 | 131 | 115 | 117 | 114 | 115
Percentage of participants
  Redness: Mild | 6.1 [2.7 to 11.7] | 10.7 [6.0 to 17.3] | 0.9 [0.0 to 4.7] | 4.3 [1.4 to 9.7] | 2.6 [0.5 to 7.5] | 2.6 [0.5 to 7.4]
  Redness: Moderate | 3.8 [1.3 to 8.7] | 1.5 [0.2 to 5.4] | 2.6 [0.5 to 7.4] | 3.4 [0.9 to 8.5] | 1.8 [0.2 to 6.2] | 1.7 [0.2 to 6.1]
  Redness: Severe | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Redness: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Swelling: Mild | 4.6 [1.7 to 9.7] | 9.9 [5.4 to 16.4] | 5.2 [1.9 to 11.0] | 3.4 [0.9 to 8.5] | 0.9 [0.0 to 4.8] | 8.7 [4.2 to 15.4]
  Swelling: Moderate | 5.3 [2.2 to 10.7] | 6.9 [3.2 to 12.6] | 4.3 [1.4 to 9.9] | 6.8 [3.0 to 13.0] | 4.4 [1.4 to 9.9] | 1.7 [0.2 to 6.1]
  Swelling: Severe | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Swelling: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Pain at injection site: Mild | 38.2 [29.8 to 47.1] | 33.6 [25.6 to 42.4] | 38.3 [29.4 to 47.8] | 40.2 [31.2 to 49.6] | 26.3 [18.5 to 35.4] | 41.7 [32.6 to 51.3]
  Pain at injection site: Moderate | 21.4 [14.7 to 29.4] | 29.0 [21.4 to 37.6] | 6.1 [2.5 to 12.1] | 13.7 [8.0 to 21.3] | 1.8 [0.2 to 6.2] | 8.7 [4.2 to 15.4]
  Pain at injection site: Severe | 0.8 [0.0 to 4.2] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Post vaccination 2: Redness: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Redness: Mild |  |  |  |  |  | 4.1 [1.1 to 10.1]
  Post vaccination 2: Redness: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Redness: Moderate |  |  |  |  |  | 5.1 [1.7 to 11.5]
  Post vaccination 2: Redness: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Redness: Severe |  |  |  |  |  | 1.0 [0.0 to 5.6]
  Post vaccination 2: Redness: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Redness: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Swelling: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Swelling: Mild |  |  |  |  |  | 5.1 [1.7 to 11.5]
  Post vaccination 2: Swelling: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Swelling: Moderate |  |  |  |  |  | 3.1 [0.6 to 8.7]
  Post vaccination 2: Swelling: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Swelling: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Swelling: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Swelling: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Pain at injection site: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Pain at injection site: Mild |  |  |  |  |  | 33.7 [24.4 to 43.9]
  Post vaccination 2: Pain at injection site: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Pain at injection site: Moderate |  |  |  |  |  | 8.2 [3.6 to 15.5]
  Post vaccination 2: Pain at injection site: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Pain at injection site: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Pain at injection site: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Pain at injection site: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]

22. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination for 1-Visit Schedule (Initial Enrollment): Substudy B
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, chills, new/worsened muscle pain & new /worsened joint pain & recorded by participants in electronic diary. Fever defined as oral temperature >=38.0 deg C & categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C & >40.0 deg C. Vomiting graded as: G 1: 1-2 times in 24 hrs; G 2: >2 times in 24 hrs; G 3: required IV hydration; G 4: emergency room visit/ hospitalization for hypotensive shock. Diarrhea graded as: G 1: 2-3 loose stools in 24 hrs; G 2: 4-5 loose stools in 24 hrs; G 3: 6 or more loose stools in 24 hrs & G 4: emergency room visit/ hospitalization. Headache, fatigue, chills, new/worsened muscle pain & new/worsened joint pain: G 1: didn't interfere with activity; G 2: some interference with activity; G 3: prevented daily routine activity & G 4: emergency room visit/ hospitalization. Exact 2-sided confidence interval based on Clopper and Pearson method.
Time Frame: From Day 1 to Day 7 after vaccination
Population: Safety population included all the participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) at Day 1 as part of initial enrollment.
Arm/Group | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 14 | 16 | 15
Percentage of participants
  Fever: >=38.0 degree C to 38.4 degree C | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 6.3 [0.2 to 30.2] | 13.3 [1.7 to 40.5]
  Fever: >38.4 degree C to 38.9 degree C | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Fever: >38.9 degree C to 40.0 degree C | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Fever: >40.0 degree C | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Fatigue: Mild | 12.5 [1.6 to 38.3] | 13.3 [1.7 to 40.5] | 12.5 [1.6 to 38.3] | 26.7 [7.8 to 55.1] | 0.0 [0.0 to 23.2] | 18.8 [4.0 to 45.6] | 13.3 [1.7 to 40.5]
  Fatigue: Moderate | 18.8 [4.0 to 45.6] | 20.0 [4.3 to 48.1] | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9] | 21.4 [4.7 to 50.8] | 6.3 [0.2 to 30.2] | 13.3 [1.7 to 40.5]
  Fatigue: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Fatigue: grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Headache: Mild | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9] | 18.8 [4.0 to 45.6] | 13.3 [1.7 to 40.5] | 14.3 [1.8 to 42.8] | 6.3 [0.2 to 30.2] | 20.0 [4.3 to 48.1]
  Headache: Moderate | 18.8 [4.0 to 45.6] | 13.3 [1.7 to 40.5] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Headache: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Headache: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Chills: Mild | 12.5 [1.6 to 38.3] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9]
  Chills: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9]
  Chills: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Chills: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Vomiting: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Vomiting: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Vomiting: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Vomiting: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Diarrhea: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9]
  Diarrhea: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8]
  Diarrhea: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  Diarrhea: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  New or worsened muscle pain: Mild | 12.5 [1.6 to 38.3] | 13.3 [1.7 to 40.5] | 18.8 [4.0 to 45.6] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 23.2] | 6.3 [0.2 to 30.2] | 20.0 [4.3 to 48.1]
  New or worsened muscle pain: Moderate | 12.5 [1.6 to 38.3] | 6.7 [0.2 to 31.9] | 12.5 [1.6 to 38.3] | 0.0 [0.0 to 21.8] | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  New or worsened muscle pain: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  New or worsened joint pain: Mild | 6.3 [0.2 to 30.2] | 13.3 [1.7 to 40.5] | 6.3 [0.2 to 30.2] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 13.3 [1.7 to 40.5]
  New or worsened joint pain: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 20.6] | 6.7 [0.2 to 31.9]
  New or worsened joint pain: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 21.8]

23. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination 1 for 2- Visit Schedule (Initial Enrollment): Substudy B
Description: as for outcome 22
Time Frame: From Day 1 to Day 7 after vaccination 1
Population: Safety population included all the participants who received the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding AA strains at dose level combination 1 administered 21 days apart as part of initial enrollment.
- SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding AA strains at dose level combination 2 administered 21 days apart as part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16
Percentage of participants
  Fever: >=38.0 degree C to 38.4°C | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Fever: >38.4 degree C to 38.9 degree C | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Fever: >38.9 degree C to 40.0 degree C | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Fever: >40.0 degree C | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Fatigue: Mild | 14.3 [1.8 to 42.8] | 40.0 [16.3 to 67.7] | 0.0 [0.0 to 20.6] | 31.3 [11.0 to 58.7]
  Fatigue: Moderate | 21.4 [4.7 to 50.8] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 20.6]
  Fatigue: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Fatigue: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Headache: Mild | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5] | 6.3 [0.2 to 30.2] | 12.5 [1.6 to 38.3]
  Headache: Moderate | 28.6 [8.4 to 58.1] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Headache: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Headache: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Chills: Mild | 14.3 [1.8 to 42.8] | 20.0 [4.3 to 48.1] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 20.6]
  Chills: Moderate | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Chills: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Chills: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Vomiting: Mild | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Vomiting: Moderate | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Vomiting: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Vomiting: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Diarrhea: Mild | 21.4 [4.7 to 50.8] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Diarrhea: Moderate | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Diarrhea: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  Diarrhea: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Mild | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Moderate | 14.3 [1.8 to 42.8] | 6.7 [0.20 to 31.9] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened joint pain: Mild | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 30.2]
  New or worsened joint pain: Moderate | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 6.3 [0.2 to 30.2]
  New or worsened joint pain: Severe | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6]

24. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination 2 for 2-Visit Schedule (Initial Enrollment) : Substudy B
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, chills, new/worsened muscle pain & new /worsened joint pain & recorded by participants in electronic diary. Fever defined as oral temperature >=38.0 deg C & categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C & >40.0 deg C. Vomiting graded as: G 1: 1-2 times in 24 hrs; G 2: >2 times in 24 hrs; G 3: required IV hydration; G 4: emergency room visit/ hospitalization for hypotensive shock. Diarrhea graded as: G: 1: 2-3 loose stools in 24 hrs; G 2: 4-5 loose stools in 24 hrs; G 3: 6 or more loose stools in 24 hrs & G 4: emergency room visit/ hospitalization. Headache, fatigue, chills, new/worsened muscle pain & new/worsened joint pain: G 1: didn't interfere with activity; G 2: some interference with activity; G 3: prevented daily routine activity & G 4: emergency room visit/ hospitalization. Exact 2-sided confidence interval based on Clopper and Pearson method.
Time Frame: From day 1 to day 7 of vaccination 2
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 13 | 14 | 15 | 16
Percentage of participants
  Fever: >=38.0 degree C to 38.4 degree C | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  Fever: >38.4 degree C to 38.9 degree C | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Fever: >38.9 degree C to 40.0 degree C | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Fever: >40.0 degree C | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Fatigue: Mild | 23.1 [5.0 to 53.8] | 21.4 [4.7 to 50.8] | 13.3 [1.7 to 40.5] | 12.5 [1.6 to 38.3]
  Fatigue: Moderate | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5] | 6.3 [0.2 to 30.2]
  Fatigue: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Fatigue: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Headache: Mild | 7.7 [0.2 to 36.0] | 14.3 [1.8 to 42.8] | 26.7 [7.8 to 55.1] | 12.5 [1.6 to 38.3]
  Headache: Moderate | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Headache: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Headache: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Chills: Mild | 15.4 [1.9 to 45.4] | 14.3 [1.8 to 42.8] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  Chills: Moderate | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  Chills: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Chills: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Vomiting: Mild | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Vomiting: Moderate | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 6.3 [0.2 to 30.2]
  Vomiting: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Vomiting: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Diarrhea: Mild | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Diarrhea: Moderate | 0.0 [0.0 to 24.7] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Diarrhea: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  Diarrhea: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Mild | 23.1 [5.0 to 53.8] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8] | 12.5 [1.6 to 38.3]
  New or worsened muscle pain: Moderate | 0.0 [0.0 to 24.7] | 7.1 [0.2 to 33.9] | 6.7 [0.2 to 31.9] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  New or worsened joint pain: Mild | 7.7 [0.2 to 36.0] | 14.3 [1.8 to 42.8] | 6.7 [0.2 to 31.9] | 12.5 [1.6 to 38.3]
  New or worsened joint pain: Moderate | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  New or worsened joint pain: Severe | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6]

25. Primary Outcome: Percentage of Participants Reporting Systemic Events After Vaccination for Expanded Enrollment: Substudy B
Description: as for outcome 22
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment: Participants aged 18 to 64 years received a single intramuscular injection of qIRV dose level 2 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 131 | 131 | 115 | 117 | 114 | 115
Percentage of participants
  Fever: >=38.0 degree C to 38.4 degree C | 3.1 [0.8 to 7.6] | 5.3 [2.2 to 10.7] | 0.9 [0.0 to 4.7] | 3.4 [0.9 to 8.5] | 2.6 [0.5 to 7.5] | 0.0 [0.0 to 3.2]
  Fever: >38.4 degree C to 38.9 degree C | 0.8 [0.0 to 4.2] | 1.5 [0.2 to 5.4] | 1.7 [0.2 to 6.1] | 1.7 [0.2 to 6.0] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Fever: >38.9 degree C to 40.0 degree C | 0.0 [0.0 to 2.8] | 1.5 [0.2 to 5.4] | 0.9 [0.0 to 4.7] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Fever: >40.0 degree C | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 31.2] | 0.0 [0.0 to 3.2]
  Fatigue: Mild | 15.3 [9.6 to 22.6] | 16.8 [10.8 to 24.3] | 13.9 [8.2 to 21.6] | 21.4 [14.3 to 29.9] | 12.3 [6.9 to 19.7] | 9.6 [4.9 to 16.5]
  Fatigue: Moderate | 26.7 [19.4 to 35.2] | 22.1 [15.4 to 30.2] | 19.1 [12.4 to 27.5] | 19.7 [12.9 to 28.0] | 7.9 [3.7 to 14.5] | 8.7 [4.2 to 15.4]
  Fatigue: Severe | 1.5 [0.2 to 5.4] | 2.3 [0.5 to 6.5] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.9 [0.0 to 4.8] | 2.6 [0.5 to 7.4]
  Fatigue: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Headache: Mild | 13.0 [7.7 to 20.0] | 17.6 [11.5 to 25.2] | 15.7 [9.5 to 23.6] | 13.7 [8.0 to 21.3] | 8.8 [4.3 to 15.5] | 8.7 [4.2 to 15.4]
  Headache: Moderate | 25.2 [18.0 to 33.5] | 18.3 [12.1 to 26.0] | 4.3 [1.4 to 9.9] | 13.7 [8.0 to 21.3] | 1.8 [0.2 to 6.2] | 4.3 [1.4 to 9.9]
  Headache: Severe | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Headache: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Chills: Mild | 9.9 [5.4 to 16.4] | 9.9 [5.4 to 16.4] | 3.5 [1.0 to 8.7] | 9.4 [4.8 to 16.2] | 4.4 [1.4 to 9.9] | 7.8 [3.6 to 14.3]
  Chills: Moderate | 9.2 [4.8 to 15.5] | 9.9 [5.4 to 16.4] | 3.5 [1.0 to 8.7] | 7.7 [3.6 to 14.1] | 0.0 [0.0 to 3.2] | 4.3 [1.4 to 9.9]
  Chills: Severe | 0.0 [0.0 to 2.8] | 0.8 [0.0 to 4.2] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Chills: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Vomiting: Mild | 2.3 [0.5 to 6.5] | 1.5 [0.2 to 5.4] | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.0] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7]
  Vomiting: Moderate | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Vomiting: Severe | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Vomiting: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Diarrhea: Mild | 10.7 [6.0 to 17.3] | 5.3 [2.2 to 10.7] | 3.5 [1.0 to 8.7] | 3.4 [0.9 to 8.5] | 5.3 [2.0 to 11.1] | 3.5 [1.0 to 8.7]
  Diarrhea: Moderate | 1.5 [0.2 to 5.4] | 1.5 [0.2 to 5.4] | 0.9 [0.0 to 4.7] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.1]
  Diarrhea: Severe | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Diarrhea: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  New or worsened muscle pain: Mild | 13.0 [7.7 to 20.0] | 13.0 [7.7 to 20.0] | 8.7 [4.2 to 15.4] | 10.3 [5.4 to 17.2] | 4.4 [1.4 to 9.9] | 9.6 [4.9 to 16.5]
  New or worsened muscle pain: Moderate | 13.7 [8.4 to 20.8] | 18.3 [12.1 to 26.0] | 7.8 [3.6 to 14.3] | 11.1 [6.1 to 18.3] | 2.6 [0.5 to 7.5] | 1.7 [0.2 to 6.1]
  New or worsened muscle pain: Severe | 0.8 [0.0 to 4.2] | 0.8 [0.0 to 4.2] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.9 [0.0 to 4.8] | 0.9 [0.0 to 4.7]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  New or worsened joint pain: Mild | 8.4 [4.3 to 14.5] | 9.2 [4.8 to 15.5] | 6.1 [2.5 to 12.1] | 6.0 [2.4 to 11.9] | 0.0 [0.0 to 3.2] | 2.6 [0.5 to 7.4]
  New or worsened joint pain: Moderate | 9.2 [4.8 to 15.5] | 8.4 [4.3 to 14.5] | 7.0 [3.1 to 13.2] | 11.1 [6.1 to 18.3] | 0.9 [0.0 to 4.8] | 2.6 [0.5 to 7.4]
  New or worsened joint pain: Severe | 0.8 [0.0 to 4.2] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 2.8] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2]
  Post vaccination 2: Fever: >=38.0 degree C to 38.4 degree C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fever: >=38.0 degree C to 38.4 degree C |  |  |  |  |  | 2.0 [0.2 to 7.2]
  Post vaccination 2: Fever: >38.4 degree C to 38.9 degree C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fever: >38.4 degree C to 38.9 degree C |  |  |  |  |  | 3.1 [0.6 to 8.7]
  Post vaccination 2: Fever: >38.9 degree C to 40.0 degree C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fever: >38.9 degree C to 40.0 degree C |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Fever: >40.0 degree C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fever: >40.0 degree C |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Fatigue: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fatigue: Mild |  |  |  |  |  | 11.2 [5.7 to 19.2]
  Post vaccination 2: Fatigue: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fatigue: Moderate |  |  |  |  |  | 17.3 [10.4 to 26.3]
  Post vaccination 2: Fatigue: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fatigue: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Fatigue: grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Fatigue: grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Headache: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Headache: Mild |  |  |  |  |  | 12.2 [6.5 to 20.4]
  Post vaccination 2: Headache: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Headache: Moderate |  |  |  |  |  | 12.2 [6.5 to 20.4]
  Post vaccination 2: Headache: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Headache: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Headache: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Headache: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Chills: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Chills: Mild |  |  |  |  |  | 8.2 [3.6 to 15.5]
  Post vaccination 2: Chills: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Chills: Moderate |  |  |  |  |  | 6.1 [2.3 to 12.9]
  Post vaccination 2: Chills: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Chills: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Chills: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Chills: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Vomiting: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Vomiting: Mild |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Vomiting: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Vomiting: Moderate |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Vomiting: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Vomiting: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Vomiting: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Vomiting: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Diarrhea: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Diarrhea: Mild |  |  |  |  |  | 2.0 [0.2 to 7.2]
  Post vaccination 2: Diarrhea: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Diarrhea: Moderate |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Diarrhea: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Diarrhea: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: Diarrhea: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: Diarrhea: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: New or worsened muscle pain: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened muscle pain: Mild |  |  |  |  |  | 6.1 [2.3 to 12.9]
  Post vaccination 2: New or worsened muscle pain: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened muscle pain: Moderate |  |  |  |  |  | 6.1 [2.3 to 12.9]
  Post vaccination 2: New or worsened muscle pain: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened muscle pain: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: New or worsened muscle pain: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened muscle pain: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: New or worsened joint pain: Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened joint pain: Mild |  |  |  |  |  | 4.1 [1.1 to 10.1]
  Post vaccination 2: New or worsened joint pain: Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened joint pain: Moderate |  |  |  |  |  | 4.1 [1.1 to 10.1]
  Post vaccination 2: New or worsened joint pain: Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened joint pain: Severe |  |  |  |  |  | 0.0 [0.0 to 3.7]
  Post vaccination 2: New or worsened joint pain: Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 115
  Post vaccination 2: New or worsened joint pain: Grade 4 |  |  |  |  |  | 0.0 [0.0 to 3.7]

26. Primary Outcome: Percentage of Participants Reporting Adverse Events From First Vaccination Until 4 Weeks After Last Vaccination: Substudy B
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Only AEs collected by non-systematic assessment (i.e, excluding local reactions and systematic events) were reported in this outcome measure.
Time Frame: From first vaccination to 4 weeks after last vaccination (i.e., Vaccination 1 for 1-visit schedule arms and Vaccination 2 for 2-visit schedule arms)
Population: Safety population included all the participants who received the study intervention.
Measure: Number; unit: Percentage of participants
Groups:
- SSB: Licensed QIV+bIRV AA (Dose Level Combination 1): 1-Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of qIRV dose level 2, dose combination 2 administered at day 1 as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) as a part of expanded enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV+bIRV AA (Dose Level Combination 1): 1-Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 14 | 15 | 15 | 131 | 131 | 116 | 117 | 115 | 117
Percentage of participants | 7.1 | 13.3 | 6.3 | 6.3 | 12.5 | 0 | 6.3 | 0 | 0 | 0 | 0 | 1.5 | 3.1 | 6.9 | 8.5 | 7.0 | 12.0

27. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events From First Vaccination Until 6 Months After Last Vaccination: Substudy B
Description: as for outcome 7
Time Frame: From first vaccination to 6 month after last vaccination (i.e., Vaccination 1 for 1-visit schedule arms and Vaccination 2 for 2-visit schedule arms)
Population: Safety population included all the participants who received the study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: Licensed QIV+bIRV AA (Dose Level Combination 2): 1-Visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 2) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, dose combination 1 as a part of expanded enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV+bIRV AA (Dose Level Combination 1): 1-Visit Schedule: Initial Enrollment | SSB: Licensed QIV+bIRV AA (Dose Level Combination 2): 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 16 | 14 | 15 | 15 | 131 | 131 | 116 | 117 | 115 | 117
Percentage of participants | 0.00 [0.0 to 21.8] | 0.00 [0.0 to 23.2] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 20.6] | 0 [0 to 0] | 0 [0 to 0] | 0.0 [0.0 to 21.8] | 0 [0 to 0] | 0.0 [0.0 to 2.8] | 1.5 [0.2 to 5.4] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0 [0 to 0]

28. Primary Outcome: Percentage of Participants Reporting Abnormal Troponin I Laboratory Values 2 Days After Vaccination 1 for 2-Visit Schedule (Initial Enrollment): Substudy B
Description: Percentage of participants reporting abnormal troponin I laboratory values 2 days after vaccination 1 were reported in this outcome measure.
Time Frame: 2 days after vaccination 1
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16
Percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

29. Primary Outcome: Percentage of Participants Reporting Abnormal Troponin I Laboratory Values 2 Days After Vaccination 2 for 2-Visit Schedule (Initial Enrollment): Substudy B
Description: Percentage of participants reporting abnormal troponin I laboratory values 2 days after vaccination 2 were reported in this outcome measure.
Time Frame: 2 days after vaccination 2
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16
Percentage of participants | 0 | 0 | 0 | 0

30. Primary Outcome: Percentage of Participants Reporting Abnormal Troponin I Laboratory Values 2 Days After Vaccination for 1-Visit Schedule (Initial Enrollment): Substudy B
Description: Percentage of participants reporting abnormal troponin I laboratory values 2 days after vaccination were reported in this outcome measure.
Time Frame: 2 days after vaccination
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 16 | 15 | 16 | 15 | 14 | 16 | 15
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Primary Outcome: Percentage of Participants Reporting Abnormal Troponin I Laboratory Values 2 Days After Vaccination for Expanded Enrollment: Substudy B
Description: as for outcome 30
Time Frame: 2 days after last vaccination (i.e., Vaccination 1 for 1-visit schedule arms and Vaccination 2 for 2-visit schedule arms)
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 131 | 131 | 115 | 117 | 114 | 115
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

32. Primary Outcome: Percentage of Participants Reporting New ECG Abnormalities 2 Days After Vaccination 1 for 2-Visit Schedule (Initial Enrollment): Substudy B
Description: Twelve lead ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position. An ECG abnormality was defined as any new abnormality that, as judged by a cardiologist, was consistent with probable or possible myocarditis or pericarditis, including: Sustained atrial or ventricular arrhythmias, Second-degree Mobitz Type II or worse atrioventricular block, new bundle branch block and Diffuse ST-segment elevation or PR-segment inversion, compatible with pericarditis.
Time Frame: 2 days after vaccination 1
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Groups:
- SSB: QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV dose level combination 2 administered 21 days apart as a part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 13 | 14 | 16 | 16
Percentage of participants | 0 | 0 | 0 | 0

33. Primary Outcome: Percentage of Participants Reporting New ECG Abnormalities 2 Days After Vaccination 2 for 2-Visit Schedule (Initial Enrollment): Substudy B
Description: as for outcome 32
Time Frame: 2 days after vaccination 2
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Groups:
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV encoding AA strains at dose Level combination 2 administered 21 days apart as a part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment
Number analyzed (Participants) | 13 | 14 | 16 | 16
Percentage of participants | 0 | 0 | 0 | 0

34. Primary Outcome: Percentage of Participants Reporting New ECG Abnormalities 2 Days After Vaccination 1 for 1-Visit Schedule (Initial Enrollment): Substudy B
Description: as for outcome 32
Time Frame: 2 days after vaccination 1
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 16 | 15 | 16 | 16 | 14 | 15 | 15
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Primary Outcome: Percentage of Participants Reporting New ECG Abnormalities 2 Days After Vaccination for Expanded Enrollment: Substudy B
Description: as for outcome 32
Time Frame: as for outcome 31
Population: as for outcome 27
Measure: Number; unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 131 | 131 | 115 | 117 | 114 | 115
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HAI) Titers at Weeks 1, 4 and 8 After Vaccination 1: Substudy A
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLQ.
Time Frame: Weeks 1, 4 and 8 after vaccination 1
Population: Vaccination 1 evaluable immunogenicity population (EIP) included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame (26-35 days) after vaccination 1; had at least 1 valid and determinate assay result at the 4-week post-vaccination 1 visit and had no major protocol deviations before vaccination 2. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
Titers
  1 Week after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 12 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: A1 | 51.5 [20.6 to 128.4] | 80.0 [28.6 to 223.8] | 63.5 [21.2 to 190.4] | 80.0 [28.7 to 223.2] | 40.0 [20.9 to 76.7] |  |  |  |  |  | 80.0 [44.4 to 144.2] | 115.8 [73.4 to 182.6] | 75.5 [33.0 to 172.9] | 68.2 [43.2 to 107.7] | 127.0 [69.4 to 232.2] | 69.0 [39.9 to 119.3] | 100.8 [47.0 to 216.2]
  1 Week after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: B1 |  |  |  |  |  | 37.9 [22.4 to 64.2] | 22.3 [12.7 to 39.1] | 29.2 [17.3 to 49.4] | 56.6 [37.6 to 85.1] | 29.2 [14.9 to 57.1] | 35.3 [19.0 to 65.4] | 24.1 [15.4 to 37.6] | 20.0 [10.7 to 37.3] | 32.3 [20.3 to 51.4] | 42.4 [26.3 to 68.3] | 19.0 [10.7 to 33.9] | 17.4 [11.0 to 27.7]
  4 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: A1 | 109.6 [41.9 to 287.0] | 205.4 [65.0 to 649.2] | 186.6 [98.4 to 354.1] | 314.0 [117.2 to 841.1] | 122.6 [56.5 to 266.0] |  |  |  |  |  | 287.9 [120.3 to 689.1] | 192.5 [120.4 to 307.8] | 137.1 [66.4 to 283.0] | 129.3 [70.8 to 236.0] | 134.5 [68.1 to 265.7] | 176.7 [84.8 to 368.0] | 204.6 [106.0 to 395.1]
  4 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: B1 |  |  |  |  |  | 69.0 [41.8 to 113.8] | 37.9 [21.8 to 65.9] | 66.2 [27.3 to 160.6] | 72.5 [41.3 to 127.2] | 22.7 [12.2 to 42.1] | 66.2 [31.2 to 140.7] | 31.7 [18.9 to 53.2] | 33.6 [19.7 to 57.4] | 40.0 [23.9 to 66.8] | 31.7 [15.6 to 64.6] | 21.0 [11.1 to 39.7] | 21.9 [11.5 to 41.9]
  8 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 10 | 15 | 12 | 13 | 12 | 13 | 15
  8 Weeks after Vaccination 1: A1 | 70.5 [30.0 to 165.7] | 137.1 [46.2 to 406.7] | 117.6 [52.6 to 262.8] | 162.8 [64.5 to 411.0] | 68.2 [34.3 to 135.6] |  |  |  |  |  | 197.0 [61.1 to 634.6] | 115.8 [68.8 to 194.8] | 108.8 [42.6 to 278.1] | 89.0 [50.7 to 156.3] | 95.1 [57.6 to 157.1] | 104.4 [46.4 to 235.2] | 133.0 [71.3 to 248.1]
  8 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 10 | 15 | 12 | 13 | 12 | 13 | 15
  8 Weeks after Vaccination 1: B1 |  |  |  |  |  | 48.8 [30.1 to 79.0] | 27.5 [13.4 to 56.4] | 42.6 [15.2 to 119.3] | 46.4 [26.2 to 82.0] | 20.0 [11.5 to 34.7] | 37.3 [16.9 to 82.3] | 17.4 [9.9 to 30.7] | 17.8 [8.9 to 35.8] | 27.5 [16.2 to 46.8] | 22.4 [12.8 to 39.2] | 16.2 [9.3 to 28.0] | 20.0 [11.9 to 33.7]
  1 Week after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 160.0 [112.6 to 227.3] | 87.7 [49.2 to 156.4]
  4 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 88.3 [51.4 to 151.7] | 57.9 [43.5 to 77.0]
  8 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 84.4 [52.9 to 134.6] | 45.9 [30.3 to 69.6]
  1 Week after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 12.8 [8.3 to 19.7] | 24.1 [15.4 to 37.6]
  4 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 17.2 [9.8 to 30.5] | 31.7 [17.9 to 56.4]
  8 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 14.5 [8.8 to 24.0] | 23.0 [14.5 to 36.5]

37. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in HAI Titers From Before Vaccination to 1, 4, and 8 Weeks After Vaccination 1: Substudy A
Description: Geometric mean fold rise (GMFR) was defined as ratios of the results after vaccination to the results before vaccination. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. When prevaccination assay results were lower than the LLOQ and the postvaccination results were greater than or equal to the LLOQ, the prevaccination assay results were set to LLOQ for the GMFR calculation.
Time Frame: Before vaccination to 1, 4 and 8 weeks after vaccination 1
Population: Vaccination 1 evaluable immunogenicity population included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame (26-35 days) after vaccination 1; had at least 1 valid and determinate assay result at the 4-week post-vaccination 1 visit and had no major protocol deviations before vaccination 2. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
Fold Rise
  1 Week after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 12 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: A1 | 2.3 [1.4 to 3.7] | 2.7 [1.6 to 4.5] | 2.2 [1.2 to 3.8] | 4.7 [2.3 to 9.7] | 2.4 [1.3 to 4.3] |  |  |  |  |  | 5.5 [3.0 to 10.0] | 4.0 [2.2 to 7.1] | 3.4 [2.0 to 5.6] | 3.8 [2.6 to 5.4] | 4.0 [2.1 to 7.7] | 4.4 [2.8 to 6.9] | 4.8 [2.4 to 9.7]
  1 Week after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 11 | 14 | 10 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: B1 |  |  |  |  |  | 1.8 [1.3 to 2.5] | 1.4 [1.0 to 1.8] | 1.8 [1.2 to 2.6] | 3.0 [1.9 to 4.7] | 2.1 [0.9 to 5.1] | 2.0 [1.2 to 3.3] | 1.9 [1.5 to 2.5] | 1.8 [1.2 to 2.7] | 1.7 [1.3 to 2.2] | 2.2 [1.3 to 3.9] | 1.6 [1.1 to 2.3] | 1.6 [1.1 to 2.3]
  1 Week after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.2 [1.0 to 1.6] | 1.6 [1.3 to 2.0]
  1 Week after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.6 [1.6 to 4.1] | 1.4 [1.0 to 2.0]
  4 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: A1 | 4.0 [1.8 to 9.0] | 5.4 [3.0 to 9.8] | 4.0 [2.1 to 7.7] | 12.7 [6.6 to 24.4] | 3.8 [1.9 to 7.4] |  |  |  |  |  | 17.4 [6.4 to 47.0] | 6.3 [3.5 to 11.5] | 6.5 [4.6 to 9.0] | 6.5 [3.2 to 13.2] | 4.5 [2.2 to 9.0] | 8.8 [5.4 to 14.5] | 7.4 [3.2 to 17.1]
  4 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: B1 |  |  |  |  |  | 3.6 [2.4 to 5.5] | 2.2 [1.7 to 3.0] | 4.5 [2.2 to 9.6] | 3.8 [2.5 to 5.8] | 2.1 [1.0 to 4.4] | 3.5 [1.6 to 7.6] | 2.2 [1.6 to 3.0] | 2.4 [1.4 to 4.1] | 1.9 [1.0 to 3.5] | 1.9 [1.1 to 3.2] | 1.7 [1.3 to 2.3] | 1.9 [1.2 to 3.1]
  4 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.6 [1.1 to 2.4] | 1.8 [1.3 to 2.6]
  4 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.6 [2.6 to 8.4] | 2.3 [1.6 to 3.3]
  8 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 10 | 15 | 12 | 13 | 12 | 14 | 15
  8 Weeks after Vaccination 1: A1 | 2.7 [1.4 to 5.2] | 3.8 [2.0 to 7.3] | 4.0 [2.1 to 7.7] | 7.7 [4.1 to 14.7] | 3.1 [1.3 to 7.4] |  |  |  |  |  | 13.0 [3.4 to 49.8] | 4.0 [2.3 to 7.0] | 4.8 [3.0 to 7.9] | 5.2 [2.8 to 9.8] | 3.0 [1.5 to 5.8] | 5.2 [3.2 to 8.6] | 5.5 [2.5 to 12.4]
  8 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 10 | 15 | 12 | 13 | 12 | 14 | 15
  8 Weeks after Vaccination 1: B1 |  |  |  |  |  | 2.6 [1.8 to 3.7] | 2.1 [1.4 to 3.3] | 2.9 [1.3 to 6.4] | 2.4 [1.6 to 3.6] | 1.6 [0.8 to 3.4] | 2.8 [1.2 to 6.4] | 1.7 [1.1 to 2.4] | 1.7 [1.0 to 2.8] | 1.7 [1.1 to 2.7] | 1.4 [0.9 to 2.3] | 1.4 [1.1 to 1.7] | 1.9 [1.3 to 2.9]
  8 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.4 [0.9 to 2.1] | 1.4 [1.1 to 1.9]
  8 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.3 [1.0 to 5.5] | 1.2 [0.7 to 2.0]

38. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for Each Strain At 1, 4, and 8 Weeks After Vaccination 1: Substudy A
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: At 1, 4 and 8 Weeks after vaccination 1
Population: Vaccination 1 EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame (26-35 days) after Vaccination 1; had at least 1 valid and determinate assay result at the 4-week post-vaccination 1 visit and had no major protocol deviations before Vaccination 2. Here, 'Number Analyzed' signifies number of participants evaluable for the specified row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 14 | 13 | 11 | 14 | 10 | 11 | 15 | 12 | 13 | 12 | 14 | 15
Percentage of participants
  1 Week after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 12 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: A1 | 45.5 [16.7 to 76.6] | 33.3 [9.9 to 65.1] | 33.3 [7.5 to 70.1] | 69.2 [38.6 to 90.9] | 50.0 [21.1 to 78.9] |  |  |  |  |  | 90.9 [58.7 to 99.8] | 60.0 [32.3 to 83.7] | 50.0 [21.1 to 78.9] | 76.9 [46.2 to 95.0] | 66.7 [34.9 to 90.1] | 71.4 [41.9 to 91.6] | 46.7 [21.3 to 73.4]
  1 Week after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 11 | 14 | 10 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: B1 |  |  |  |  |  | 7.7 [0.2 to 36.0] | 7.7 [0.2 to 36.0] | 27.3 [6.0 to 61.0] | 42.9 [17.7 to 71.1] | 40.0 [12.2 to 73.8] | 18.2 [2.3 to 51.8] | 20.0 [4.3 to 48.1] | 16.7 [2.1 to 48.4] | 7.7 [0.2 to 36.0] | 25.0 [5.5 to 57.2] | 7.1 [0.2 to 33.9] | 13.3 [1.7 to 40.5]
  1 Week after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8]
  1 Week after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 42.9 [17.7 to 71.1] | 13.3 [1.7 to 40.5]
  4 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: A1 | 45.5 [16.7 to 76.6] | 75.0 [42.8 to 94.5] | 66.7 [29.9 to 92.5] | 92.3 [64.0 to 99.8] | 53.8 [25.1 to 80.8] |  |  |  |  |  | 90.9 [58.7 to 99.8] | 86.7 [59.5 to 98.3] | 100.0 [73.5 to 100.0] | 76.9 [46.2 to 95.0] | 66.7 [34.9 to 90.1] | 92.9 [66.1 to 99.8] | 66.7 [38.4 to 88.2]
  4 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 10 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: B1 |  |  |  |  |  | 78.6 [49.2 to 95.3] | 30.8 [9.1 to 61.4] | 63.6 [30.8 to 89.1] | 64.3 [35.1 to 87.2] | 30.0 [6.7 to 65.2] | 45.5 [16.7 to 76.6] | 40.0 [16.3 to 67.7] | 41.7 [15.2 to 72.3] | 30.8 [9.1 to 61.4] | 16.7 [2.1 to 48.4] | 14.3 [1.8 to 42.8] | 26.7 [7.8 to 55.1]
  4 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 21.4 [4.7 to 50.8] | 20.0 [4.3 to 48.1]
  4 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 57.1 [28.9 to 82.3] | 40.0 [16.3 to 67.7]
  8 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 10 | 15 | 12 | 13 | 12 | 13 | 15
  8 Weeks after Vaccination 1: A1 | 36.4 [10.9 to 69.2] | 58.3 [27.7 to 84.8] | 66.7 [29.9 to 92.5] | 84.6 [54.6 to 98.1] | 69.2 [38.6 to 90.9] |  |  |  |  |  | 70.0 [34.8 to 93.3] | 66.7 [38.4 to 88.2] | 75.0 [42.8 to 94.5] | 76.9 [46.2 to 95.0] | 50.0 [21.1 to 78.9] | 76.9 [46.2 to 95.0] | 60.0 [32.3 to 83.7]
  8 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 10 | 10 | 15 | 12 | 13 | 12 | 13 | 15
  8 Weeks after Vaccination 1: B1 |  |  |  |  |  | 35.7 [12.8 to 64.9] | 38.5 [13.9 to 68.4] | 45.5 [16.7 to 76.6] | 35.7 [12.8 to 64.9] | 20.0 [2.5 to 55.6] | 40.0 [12.2 to 73.8] | 20.0 [4.3 to 48.1] | 16.7 [2.1 to 48.4] | 7.7 [0.2 to 36.0] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 24.7] | 26.7 [7.8 to 55.1]
  8 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 46.2 [19.2 to 74.9] | 20.0 [4.3 to 48.1]
  8 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15
  8 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 7.7 [0.2 to 36.0] | 6.7 [0.2 to 31.9]

39. Secondary Outcome: Percentage of Participants With HAI Titer >=1:40 for Each Strain Before Vaccination 1 and at 1, 4, and 8 Weeks After Vaccination 1: Substudy A
Description: Percentage of participants with HAI titer >=1:40 for each strain before vaccination 1 and at 1, 4 and 8 weeks after vaccination 1 is presented in this outcome measure. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination 1 on day 1 and 1, 4 and 8 weeks after vaccination 1
Population: Vaccination 1 EIP=all eligible participants who received vaccination (vax) 1; had blood drawn for assay testing within specified time frame (26-35 days) after vax 1; had at least 1 valid and determinate assay result at 4-week post-vax 1 visit and had no major protocol deviations before vax 2. Number Analyzed=number of participants evaluable for specified rows and all participants in 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
Percentage of participants
  Prior to Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  Prior to Vaccination 1: A1 | 54.5 [23.4 to 83.3] | 50.0 [21.1 to 78.9] | 55.6 [21.2 to 86.3] | 38.5 [13.9 to 68.4] | 46.2 [19.2 to 74.9] |  |  |  |  |  | 18.2 [2.3 to 51.8] | 53.3 [26.6 to 78.7] | 33.3 [9.9 to 65.1] | 30.8 [9.1 to 61.4] | 58.3 [27.7 to 84.8] | 42.9 [17.7 to 71.1] | 40.0 [16.3 to 67.7]
  Prior to Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  Prior to Vaccination 1: B1 |  |  |  |  |  | 28.6 [8.4 to 58.1] | 15.4 [1.9 to 45.4] | 18.2 [2.3 to 51.8] | 35.7 [12.8 to 64.9] | 10.0 [0.3 to 44.5] | 27.3 [6.0 to 61.0] | 13.3 [1.7 to 40.5] | 16.7 [2.1 to 48.4] | 15.4 [1.9 to 45.4] | 8.3 [0.2 to 38.5] | 28.6 [8.4 to 58.1] | 6.7 [0.2 to 31.9]
  Prior to Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  Prior to Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 7.1 [0.2 to 33.9] | 26.7 [7.8 to 55.1]
  Prior to Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 11
  Prior to Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 64.3 [35.1 to 87.2] | 73.3 [44.9 to 92.2]
  1 Week after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: A1 | 81.8 [48.2 to 97.7] | 75.0 [42.8 to 94.5] | 66.7 [29.9 to 92.5] | 76.9 [46.2 to 95.0] | 58.3 [27.7 to 84.8] |  |  |  |  |  | 100.0 [71.5 to 100.0] | 100.0 [78.2 to 100.0] | 83.3 [51.6 to 97.9] | 92.3 [64.0 to 99.8] | 100.0 [73.5 to 100.0] | 78.6 [49.2 to 95.3] | 80.0 [51.9 to 95.7]
  1 Week after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  1 Week after Vaccination 1: B1 |  |  |  |  |  | 61.5 [31.6 to 86.1] | 30.8 [9.1 to 61.4] | 54.5 [23.4 to 83.3] | 85.7 [57.2 to 98.2] | 36.4 [10.9 to 69.2] | 54.5 [23.4 to 83.3] | 33.3 [11.8 to 61.6] | 33.3 [9.9 to 65.1] | 46.2 [19.2 to 74.9] | 66.7 [34.9 to 90.1] | 28.6 [8.4 to 58.1] | 20.0 [4.3 to 48.1]
  1 Week after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 7.1 [0.2 to 33.9] | 26.7 [7.8 to 55.1]
  1 Week after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  1 Week after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 100.0 [76.8 to 100.0] | 93.3 [68.1 to 99.8]
  4 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: A1 | 81.8 [48.2 to 97.7] | 83.3 [51.6 to 97.9] | 100.0 [66.4 to 100.0] | 92.3 [64.0 to 99.8] | 92.3 [64.0 to 99.8] |  |  |  |  |  | 100.0 [71.5 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [73.5 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [73.5 to 100.0] | 92.9 [66.1 to 99.8] | 93.3 [68.1 to 99.8]
  4 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  4 Weeks after Vaccination 1: B1 |  |  |  |  |  | 92.9 [66.1 to 99.8] | 61.5 [31.6 to 86.1] | 81.8 [48.2 to 97.7] | 85.7 [57.2 to 98.2] | 27.3 [6.0 to 61.0] | 72.7 [39.0 to 94.0] | 60.0 [32.3 to 83.7] | 66.7 [34.9 to 90.1] | 61.5 [31.6 to 86.1] | 41.7 [15.2 to 72.3] | 35.7 [12.8 to 64.9] | 40.0 [16.3 to 67.7]
  4 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 35.7 [12.8 to 64.9] | 53.3 [26.6 to 78.7]
  4 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  4 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 92.9 [66.1 to 99.8] | 93.3 [68.1 to 99.8]
  8 Weeks after Vaccination 1: A1: number analyzed (Participants) | 11 | 12 | 9 | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  8 Weeks after Vaccination 1: A1 | 81.8 [48.2 to 97.7] | 83.3 [51.6 to 97.9] | 88.9 [51.8 to 99.7] | 84.6 [54.6 to 98.1] | 76.9 [46.2 to 95.0] |  |  |  |  |  | 90.0 [55.5 to 99.7] | 93.3 [68.1 to 99.8] | 83.3 [51.6 to 97.9] | 100.0 [75.3 to 100.0] | 100.0 [73.5 to 100.0] | 84.6 [54.6 to 98.1] | 93.3 [68.1 to 99.8]
  8 Weeks after Vaccination 1: B1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 11 | 14 | 11 | 11 | 15 | 12 | 13 | 12 | 14 | 15
  8 Weeks after Vaccination 1: B1 |  |  |  |  |  | 78.6 [49.2 to 95.3] | 61.5 [31.6 to 86.1] | 63.6 [30.8 to 89.1] | 71.4 [41.9 to 91.6] | 27.3 [6.0 to 61.0] | 60.0 [26.2 to 87.8] | 33.3 [11.8 to 61.6] | 25.0 [5.5 to 57.2] | 38.5 [13.9 to 68.4] | 33.3 [9.9 to 65.1] | 23.1 [5.0 to 53.8] | 33.3 [11.8 to 61.6]
  8 Weeks after Vaccination 1: A2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  8 Weeks after Vaccination 1: A2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 100.0 [75.3 to 100.0] | 86.7 [59.5 to 98.3]
  8 Weeks after Vaccination 1: B2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15
  8 Weeks after Vaccination 1: B2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 15.4 [1.9 to 45.4] | 33.3 [11.8 to 61.6]

40. Secondary Outcome: Percentage of Participants Who Achieved HAI Seroconversion for All Strains at 1, 4, and 8 Weeks After Vaccination 1: qIRV Versus Licensed QIV, Substudy A
Description: as for outcome 38
Time Frame: At 1, 4, and 8 weeks After vaccination 1
Population: Vaccination 1 EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame (26-35 days) after vaccination 1; had at least 1 valid and determinate assay result at the 4-week post-vaccination 1 visit and had no major protocol deviations before vaccination 2. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: qIRV - Licensed QIV: Participants received a single injection of licensed QIV, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, the licensed QIV control group received either a single intramuscular dose of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
Arm/Group | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 14 | 15
Percentage of participants
  1 Week after Vaccination 1 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8]
  4 Weeks after Vaccination 1 | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 21.8]
  8 Weeks after Vaccination 1: number analyzed (Participants) | 13 | 15
  8 Weeks after Vaccination 1 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 21.8]

41. Secondary Outcome: Percentage of Participants With HAI Titers>=1:40 for All Strains Before Vaccination and at 1, 4, and 8 Weeks After Vaccination 1: qIRV Versus Licensed QIV, Substudy A
Description: Percentage of participants with HAI titer >=1:40 for all strains before vaccination 1 and 1, 4 and 8 weeks after vaccination 1 is presented in this outcome measure. Exact 2-sided 95% CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination 1 on day 1 and 1, 4, and 8 weeks after vaccination 1
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: qIRV B - Licensed QIV: Participants received a single injection of QIV, licensed, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, eligible participants received a single intramuscular dose of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
Arm/Group | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV B - Licensed QIV
Number analyzed (Participants) | 14 | 15
Percentage of participants
  Prior to Vaccination 1 | 0.0 [0.0 to 23.2] | 6.7 [0.2 to 31.9]
  1 Week after Vaccination 1 | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 21.8]
  4 Weeks after Vaccination 1 | 14.3 [1.8 to 42.8] | 26.7 [7.8 to 55.1]
  8 Weeks after Vaccination 1: number analyzed (Participants) | 13 | 15
  8 Weeks after Vaccination 1 | 0.0 [0.0 to 24.7] | 20.0 [4.3 to 48.1]

42. Secondary Outcome: Geometric Mean Ratio (GMR) of HAI Titers for Each Strain at 4 Weeks After Vaccination 1: qIRV Versus Licensed QIV, Substudy A
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution) and were reported in the descriptive section. GMRs were estimated by the ratio of the GMTs between vaccine groups, using licensed QIV group as reference and were reported in the statistical analysis section.
Time Frame: 4 weeks After vaccination 1
Population: Vaccination 1 EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame (26-35 days) after Vaccination 1; had at least 1 valid and determinate assay result at the 4-week post-vaccination 1 visit and had no major protocol deviations before Vaccination 2.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- SSA: qIRV - Licensed QIV: Participants received a single injection of licensed QIV, intramuscularly into the deltoid muscle at Day 1. Following unblinding at 8 weeks after vaccination 1, the licensed QIV control group received a single intramuscular dose of mIRV encoding A strain or B strain at dose level 4 (vaccination 2).
Arm/Group | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 14 | 15
Titers
  A1 | 176.7 [84.8 to 368.0] | 204.6 [106.0 to 395.1]
  A2 | 88.3 [51.4 to 151.7] | 57.9 [43.5 to 77.0]
  B1 | 21.0 [11.1 to 39.7] | 21.9 [11.5 to 41.9]
  B2 | 17.2 [9.8 to 30.5] | 31.7 [17.9 to 56.4]
Statistical Analysis 1: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: A1; Test type: Other; Geometric Mean Ratio = 0.86, 95% CI 2-sided [0.34 to 2.20] — GMRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the difference (qIRV group minus QIV group) and the corresponding CIs (based on the Student t distribution)
Statistical Analysis 2: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: A2; Test type: Other; Geometric Mean Ratio = 1.53, 95% CI 2-sided [0.86 to 2.70] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 3: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: B1; Test type: Other; Geometric Mean Ratio = 0.96, 95% CI 2-sided [0.40 to 2.28] — [estimate comment as in outcome 42, analysis 1]
Statistical Analysis 4: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: B2; Test type: Other; Geometric Mean Ratio = 0.54, 95% CI 2-sided [0.25 to 1.18] — [estimate comment as in outcome 42, analysis 1]

43. Secondary Outcome: Difference in Percentage of Participants Achieving HAI Seroconversion for Each Strain at 4 Weeks After Vaccination 1: qIRV Versus Licensed QIV, Substudy A
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Percentage of participants achieving seroconversion for each strain at 4 weeks after vaccination 1 and exact 2-sided 95% CI based on the Clopper and Pearson method is presented in the descriptive section. Difference in percentage of participants achieving HAI seroconversion for each strain at 4 weeks after vaccination 1 is presented in the statistical analysis section.
Time Frame: 4 weeks after vaccination 1
Population: as for outcome 42
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV
Number analyzed (Participants) | 14 | 15
Percentage of participants
  A1 | 92.9 [66.1 to 99.8] | 66.7 [38.4 to 88.2]
  A2 | 57.1 [28.9 to 82.3] | 40.0 [16.3 to 67.7]
  B1 | 14.3 [1.8 to 42.8] | 26.7 [7.8 to 55.1]
  B2 | 21.4 [4.7 to 50.8] | 20.0 [4.3 to 48.1]
Statistical Analysis 1: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: A1; Test type: Other; Difference in percentage of participants = 26.2, 95% CI 2-sided [-4.5 to 53.5] — Difference in percentage of participants achieving seroconversion, qIRV group - Licensed QIV group as reference, expressed as a percentage
Statistical Analysis 2: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: A2; Test type: Other; Difference in percentage of participants = 17.1, 95% CI 2-sided [-19.2 to 49.4] — [estimate comment as in outcome 43, analysis 1]
Statistical Analysis 3: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: B1; Test type: Other; Difference in percentage of participants = -12.4, 95% CI 2-sided [-41.7 to 19.1] — [estimate comment as in outcome 43, analysis 1]
Statistical Analysis 4: Comparison: SSA: qIRV (Dose Level 1) + QIV vs SSA: qIRV - Licensed QIV; Strain: B2; Test type: Other; Difference in percentage of participants = 1.4, 95% CI 2-sided [-29.2 to 32.5] — [estimate comment as in outcome 43, analysis 1]

44. Secondary Outcome: HAI GMTs Before Vaccination 1 and 2 and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85): Expanded Enrollment: Substudy B
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: Before vaccination 1, 2 and, 1, 4, and 8 weeks after the last vaccination (i.e. after vaccination 1 for 1-vist schedule arms and after vaccination 2 for 2-visit schedule arms)
Population: EIP included all eligible participants who received vaccination; had blood drawn for assay testing within the specified time frame (26-35 days) after last vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.Here,'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 105 | 110 | 108 | 25
Titers
  Prior to vaccination 1: A1: number analyzed (Participants) | 98 | 107 | 105 | 24
  Prior to vaccination 1: A1 | 26.7 [21.3 to 33.5] | 26.9 [21.1 to 34.4] | 27.3 [21.8 to 34.2] | 16.3 [10.3 to 25.9]
  Prior to vaccination 1: A2: number analyzed (Participants) | 97 | 108 | 105 | 24
  Prior to vaccination 1: A2 | 35.9 [30.0 to 43.1] | 27.9 [23.2 to 33.6] | 29.3 [24.5 to 35.1] | 10.0 [6.6 to 15.1]
  Prior to vaccination 1: B1: number analyzed (Participants) | 97 | 108 | 105 | 24
  Prior to vaccination 1: B1 | 20.3 [17.1 to 24.0] | 20.0 [16.8 to 23.8] | 20.7 [17.3 to 24.7] | 8.4 [6.1 to 11.6]
  Prior to vaccination 1: B2: number analyzed (Participants) | 98 | 108 | 105 | 24
  Prior to vaccination 1: B2 | 17.0 [14.4 to 20.0] | 17.5 [14.6 to 20.9] | 16.2 [13.8 to 19.0] | 8.4 [6.1 to 11.5]
  Prior to vaccination 2: A1: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: A1 |  |  |  | 108.5 [67.0 to 175.8]
  Prior to vaccination 2: A2: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: A2 |  |  |  | 75.7 [47.8 to 119.8]
  Prior to vaccination 2: B1: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: B1 |  |  |  | 18.4 [12.4 to 27.4]
  Prior to vaccination 2: B2: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: B2 |  |  |  | 12.5 [8.7 to 18.0]
  1 week after vaccination: A1: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 week after vaccination: A1 | 76.7 [60.5 to 97.3] | 88.2 [69.1 to 112.5] | 99.0 [77.6 to 126.3] | 151.4 [96.3 to 237.8]
  1 week after vaccination: A2: number analyzed (Participants) | 99 | 105 | 105 | 25
  1 week after vaccination: A2 | 68.1 [57.5 to 80.7] | 62.8 [51.9 to 75.9] | 59.0 [50.0 to 69.7] | 82.2 [54.2 to 124.8]
  1 week after vaccination: B1: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 week after vaccination: B1 | 30.7 [26.0 to 36.4] | 30.3 [25.0 to 36.7] | 48.9 [40.3 to 59.2] | 26.4 [18.1 to 38.5]
  1 week after vaccination: B2: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 week after vaccination: B2 | 22.7 [18.8 to 27.3] | 24.0 [19.9 to 28.8] | 44.2 [36.4 to 53.6] | 17.9 [12.0 to 26.8]
  4 weeks after vaccination: A1 | 121.0 [96.5 to 151.7] | 155.7 [122.9 to 197.2] | 126.4 [97.8 to 163.5] | 143.2 [87.4 to 234.5]
  4 weeks after vaccination: A2 | 99.7 [83.8 to 118.6] | 108.7 [95.8 to 123.4] | 69.0 [57.9 to 82.3] | 102.7 [64.4 to 163.7]
  4 weeks after vaccination: B1 | 33.0 [28.2 to 38.7] | 36.4 [30.4 to 43.5] | 57.7 [47.3 to 70.3] | 32.9 [21.7 to 50.0]
  4 weeks after vaccination: B2: number analyzed (Participants) | 103 | 110 | 107 | 25
  4 weeks after vaccination: B2 | 23.7 [19.9 to 28.1] | 26.9 [22.6 to 32.1] | 49.6 [40.3 to 61.1] | 15.6 [10.5 to 23.1]
  8 weeks after vaccination: A1: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after vaccination: A1 | 128.4 [101.8 to 161.8] | 128.3 [100.6 to 163.8] | 81.7 [62.9 to 106.1] | 157.0 [99.5 to 247.8]
  8 weeks after vaccination: A2: number analyzed (Participants) | 103 | 107 | 108 | 25
  8 weeks after vaccination: A2 | 95.5 [79.9 to 114.1] | 101.7 [84.6 to 122.1] | 34.3 [27.8 to 42.3] | 67.7 [43.3 to 105.9]
  8 weeks after vaccination: B1: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after vaccination: B1 | 20.4 [17.1 to 24.3] | 22.6 [18.2 to 28.0] | 30.0 [23.9 to 37.6] | 26.4 [18.1 to 38.5]
  8 weeks after vaccination: B2: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after vaccination: B2 | 17.5 [14.5 to 21.2] | 19.4 [16.2 to 23.2] | 32.4 [26.8 to 39.3] | 15.2 [10.7 to 21.5]

45. Secondary Outcome: HAI GMTs Before Vaccination 1 and 2, and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years of Age): Initial Enrollment: Substudy B
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5 × LLOQ.
Time Frame: Prior to vaccination 1 and 2, and at 1, 4, and 8 weeks after the last vaccination (i.e. after vaccination 1 for 1-vist schedule arms and after vaccination 2 for 2-visit schedule arms)
Population: as for outcome 44
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV dose Level combination 1 administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV dose Level combination 2 administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in theopposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as a part of initial enrollment.
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, encoding 2A strains and 2B strains (dose combination 1) as part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
Titers
  Prior to Vaccination 1: A1 | 25.2 [10.6 to 59.7] | 46.5 [17.6 to 122.5] | 27.4 [12.8 to 58.7] | 26.3 [13.1 to 53.1] | 23.4 [10.6 to 51.9] | 70.3 [29.2 to 168.8] | 27.5 [14.9 to 51.0] | 24.3 [11.3 to 52.2] | 32.3 [15.8 to 65.9] | 39.9 [14.2 to 111.9] | 50.6 [18.3 to 140.3]
  Prior to Vaccination 1: A2 | 32.1 [16.2 to 63.4] | 50.9 [37.1 to 69.9] | 26.9 [14.2 to 51.1] | 28.5 [15.9 to 51.1] | 36.6 [22.7 to 59.1] | 66.0 [35.4 to 122.9] | 35.5 [20.7 to 60.7] | 45.8 [33.5 to 62.6] | 20.1 [10.7 to 37.8] | 19.6 [10.7 to 35.8] | 21.0 [13.0 to 33.8]
  Prior to Vaccination 1: B1 | 16.5 [9.7 to 28.1] | 20.8 [14.3 to 30.3] | 24.7 [11.6 to 52.4] | 16.7 [8.8 to 31.7] | 19.3 [13.9 to 26.6] | 25.9 [15.8 to 42.4] | 13.7 [8.9 to 21.1] | 22.9 [14.8 to 35.5] | 11.0 [6.4 to 19.0] | 18.4 [9.4 to 36.0] | 13.0 [6.7 to 25.5]
  Prior to Vaccination 1: B2 | 14.5 [10.6 to 19.7] | 16.6 [9.8 to 28.2] | 13.1 [7.0 to 24.6] | 17.7 [8.4 to 37.5] | 14.4 [9.2 to 22.7] | 18.2 [11.1 to 29.7] | 9.1 [6.7 to 12.3] | 12.5 [9.8 to 16.1] | 10.5 [6.1 to 18.3] | 11.6 [7.1 to 18.8] | 15.7 [7.8 to 31.5]
  Prior to Vaccination 2: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A1 | 394.0 [164.0 to 946.2] | 298.6 [145.5 to 612.5] | 219.3 [99.6 to 482.7] | 160.0 [70.6 to 362.8] |  |  |  |  |  |  |
  Prior to Vaccination 2: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A2 | 149.3 [75.7 to 294.5] | 69.6 [32.3 to 150.1] | 66.2 [35.3 to 124.1] | 95.1 [55.7 to 162.5] |  |  |  |  |  |  |
  Prior to Vaccination 2: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B1 | 34.8 [18.9 to 64.1] | 42.9 [22.7 to 81.1] | 75.1 [38.3 to 147.3] | 63.5 [41.2 to 98.0] |  |  |  |  |  |  |
  Prior to Vaccination 2: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B2 | 23.0 [13.1 to 40.3] | 42.9 [20.1 to 91.3] | 33.1 [16.5 to 66.2] | 89.8 [43.6 to 185.1] |  |  |  |  |  |  |
  1 Week after last vaccination: A1 | 569.7 [291.3 to 1114.1] | 320.0 [165.2 to 619.8] | 320.0 [165.6 to 618.2] | 160.0 [77.3 to 331.1] | 151.0 [97.4 to 234.2] | 326.0 [171.5 to 619.6] | 96.2 [60.2 to 153.9] | 72.5 [35.4 to 148.4] | 134.5 [52.5 to 344.9] | 121.3 [57.2 to 257.0] | 151.0 [63.3 to 360.4]
  1 week after last vaccination: B1 | 45.9 [22.1 to 95.5] | 42.9 [24.8 to 74.0] | 66.2 [39.6 to 110.7] | 67.3 [45.9 to 98.5] | 35.6 [23.6 to 53.9] | 63.5 [29.1 to 138.8] | 18.2 [11.1 to 30.1] | 36.2 [22.7 to 57.8] | 23.5 [13.3 to 41.5] | 36.5 [20.8 to 63.8] | 28.3 [15.0 to 53.5]
  1 week after vaccination: A2 | 171.5 [90.6 to 324.6] | 113.1 [60.3 to 212.3] | 90.7 [54.9 to 150.0] | 75.5 [37.0 to 154.2] | 84.8 [54.7 to 131.4] | 151.0 [82.3 to 277.2] | 96.2 [68.6 to 135.1] | 88.3 [58.6 to 133.2] | 113.1 [56.7 to 225.6] | 45.9 [33.0 to 64.0] | 56.6 [28.4 to 112.8]
  1 week after last vaccination: B2 | 26.4 [12.5 to 55.7] | 40.0 [19.1 to 83.8] | 33.1 [16.5 to 66.2] | 75.5 [38.9 to 146.5] | 31.7 [21.5 to 46.9] | 44.9 [25.7 to 78.5] | 12.6 [8.9 to 17.8] | 25.6 [11.9 to 54.9] | 16.2 [9.6 to 27.3] | 20.0 [12.9 to 30.9] | 23.8 [11.2 to 50.6]
  4 weeks after last vaccination: A1 | 411.9 [165.5 to 1025.6] | 422.2 [225.5 to 790.6] | 320.0 [160.4 to 638.4] | 160.0 [73.8 to 347.0] | 239.7 [138.8 to 413.9] | 338.4 [179.5 to 638.0] | 335.1 [196.8 to 570.7] | 88.3 [42.4 to 184.0] | 178.0 [80.0 to 395.9] | 164.8 [81.0 to 335.6] | 332.1 [161.7 to 682.3]
  4 weeks after last vaccination: B1 | 45.9 [17.6 to 119.8] | 42.9 [26.2 to 70.2] | 58.4 [32.0 to 106.6] | 63.5 [36.9 to 109.2] | 63.5 [41.2 to 98.0] | 80.0 [35.3 to 181.4] | 38.2 [22.9 to 63.7] | 40.0 [26.4 to 60.6] | 104.4 [65.3 to 167.0] | 76.4 [56.2 to 103.8] | 151.0 [87.5 to 260.8]
  4 weeks after last vaccination: A2 | 130.0 [86.4 to 195.5] | 171.5 [99.4 to 295.9] | 124.4 [80.9 to 191.3] | 119.9 [80.6 to 178.2] | 95.1 [59.8 to 151.4] | 254.0 [171.8 to 375.5] | 145.9 [102.7 to 207.3] | 62.5 [41.7 to 93.5] | 23.5 [13.3 to 41.5] | 48.8 [26.3 to 90.3] | 37.8 [21.2 to 67.3]
  4 weeks after last vaccination: B2 | 21.4 [10.1 to 45.6] | 32.5 [16.7 to 63.1] | 22.7 [14.4 to 35.8] | 56.6 [29.1 to 109.9] | 42.4 [23.8 to 75.5] | 42.4 [23.8 to 75.5] | 18.2 [10.2 to 32.5] | 31.2 [14.6 to 67.0] | 15.3 [8.4 to 28.1] | 20.0 [12.5 to 32.0] | 26.7 [15.0 to 47.6]
  8 weeks after last vaccination: A1 | 298.6 [135.4 to 658.5] | 211.1 [130.8 to 340.9] | 170.4 [84.2 to 344.8] | 75.5 [36.1 to 158.0] | 151.0 [80.0 to 285.2] | 248.7 [104.7 to 591.0] | 175.5 [95.0 to 324.0] | 51.2 [25.6 to 102.7] | 198.0 [86.6 to 452.8] | 176.7 [86.3 to 361.8] | 370.4 [162.0 to 847.0]
  8 Week after last vaccination: B1 | 45.9 [15.8 to 133.4] | 30.3 [14.9 to 61.6] | 48.3 [28.9 to 80.8] | 44.9 [26.5 to 75.9] | 42.4 [23.8 to 75.5] | 42.6 [15.5 to 116.8] | 17.4 [9.9 to 30.7] | 23.2 [13.7 to 39.2] | 116.2 [54.5 to 247.8] | 69.0 [48.2 to 98.6] | 127.0 [79.2 to 203.7]
  8 weeks after last vaccination: A2 | 149.3 [82.5 to 270.3] | 105.6 [65.4 to 170.4] | 105.6 [65.4 to 170.4] | 63.5 [34.7 to 116.1] | 90.7 [60.4 to 136.3] | 181.5 [109.8 to 299.9] | 96.2 [47.7 to 194.4] | 31.2 [17.9 to 54.5] | 23.5 [12.3 to 44.7] | 48.8 [25.3 to 93.9] | 37.8 [19.0 to 75.2]
  8 weeks after last vaccination: B2 | 21.4 [8.8 to 52.1] | 28.3 [12.5 to 64.1] | 22.7 [10.5 to 49.2] | 56.6 [29.9 to 106.9] | 33.6 [19.7 to 57.4] | 45.4 [22.2 to 92.8] | 18.2 [9.6 to 34.8] | 23.2 [11.9 to 45.3] | 15.3 [8.2 to 28.7] | 19.0 [11.9 to 30.3] | 26.7 [14.1 to 50.4]

46. Secondary Outcome: HAI GMFR From Before Vaccination 2 to 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Expanded Enrollment: Substudy B
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5* LLOQ. When prevaccination assay results were lower than the LLOQ and the postvaccination results were greater than or equal to the LLOQ, the prevaccination assay results were set to LLOQ for the GMFR calculation.
Time Frame: From before vaccination 2 to 1, 4, and 8 weeks after the last vaccination
Population: as for outcome 44
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Groups:
- SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment: Participants aged 65-85 years received a single intramuscular injection of qIRV dose level 1 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 105 | 110 | 108 | 25
Fold Rise
  Prior to Vaccination 2: A1: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to Vaccination 2: A1 |  |  |  | 5.3 [3.4 to 8.5]
  Prior to Vaccination 2: A2: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to Vaccination 2: A2 |  |  |  | 5.5 [3.6 to 8.3]
  Prior to Vaccination 2: B1: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to Vaccination 2: B1 |  |  |  | 1.6 [1.2 to 2.2]
  Prior to Vaccination 2: B2: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to Vaccination 2: B2 |  |  |  | 1.2 [0.9 to 1.4]
  1 week after last vaccination: A1: number analyzed (Participants) | 96 | 106 | 105 | 24
  1 week after last vaccination: A1 | 2.6 [2.2 to 3.2] | 2.9 [2.4 to 3.5] | 3.3 [2.6 to 4.1] | 7.6 [4.4 to 12.8]
  1 week after last vaccination: B1: number analyzed (Participants) | 95 | 107 | 105 | 24
  1 week after last vaccination: B1 | 1.5 [1.3 to 1.6] | 1.4 [1.3 to 1.6] | 2.2 [1.8 to 2.6] | 2.2 [1.5 to 3.1]
  1 week after last vaccination: A2: number analyzed (Participants) | 94 | 105 | 105 | 25
  1 week after last vaccination: A2 | 1.8 [1.5 to 2.1] | 2.1 [1.7 to 2.5] | 1.9 [1.7 to 2.2] | 6.0 [4.0 to 9.0]
  1 week after last vaccination: B2: number analyzed (Participants) | 96 | 107 | 105 | 24
  1 week after last vaccination: B2 | 1.3 [1.2 to 1.4] | 1.3 [1.1 to 1.4] | 2.4 [1.9 to 3.0] | 1.5 [1.1 to 2.1]
  4 weeks after last vaccination: A1: number analyzed (Participants) | 98 | 107 | 105 | 24
  4 weeks after last vaccination: A1 | 4.0 [3.2 to 5.0] | 4.9 [3.9 to 6.2] | 4.1 [3.2 to 5.3] | 7.1 [4.2 to 12.2]
  4 weeks after last vaccination: B1: number analyzed (Participants) | 97 | 108 | 105 | 24
  4 weeks after last vaccination: B1 | 1.5 [1.4 to 1.7] | 1.7 [1.5 to 2.0] | 2.7 [2.2 to 3.3] | 2.7 [1.8 to 3.9]
  4 weeks after last vaccination: A2: number analyzed (Participants) | 97 | 105 | 105 | 24
  4 weeks after last vaccination: A2 | 2.6 [2.2 to 3.0] | 3.5 [3.0 to 4.0] | 2.3 [1.9 to 2.7] | 7.8 [5.1 to 11.8]
  4 weeks after last vaccination: B2: number analyzed (Participants) | 96 | 108 | 104 | 24
  4 weeks after last vaccination: B2 | 1.3 [1.2 to 1.4] | 1.4 [1.2 to 1.6] | 2.8 [2.2 to 3.5] | 1.4 [1.1 to 1.8]
  8 weeks after last vaccination: A1: number analyzed (Participants) | 98 | 106 | 105 | 24
  8 weeks after last vaccination: A1 | 4.3 [3.5 to 5.2] | 4.0 [3.2 to 5.0] | 2.7 [2.1 to 3.5] | 7.8 [4.8 to 12.8]
  8 weeks after last vaccination: A2: number analyzed (Participants) | 95 | 105 | 105 | 24
  8 weeks after last vaccination: A2 | 2.5 [2.1 to 3.0] | 3.3 [2.7 to 4.0] | 1.1 [0.9 to 1.4] | 5.0 [3.3 to 7.7]
  8 weeks after last vaccination: B1: number analyzed (Participants) | 97 | 107 | 105 | 24
  8 weeks after last vaccination: B1 | 1.0 [0.9 to 1.1] | 1.1 [0.9 to 1.3] | 1.4 [1.1 to 1.7] | 2.2 [1.6 to 3.0]
  8 weeks after last vaccination: B2: number analyzed (Participants) | 98 | 107 | 105 | 24
  8 weeks after last vaccination: B2 | 1.0 [0.8 to 1.1] | 1.0 [0.9 to 1.1] | 1.8 [1.5 to 2.2] | 1.4 [1.1 to 1.8]

47. Secondary Outcome: HAI GMFR From Before Vaccination 1 to Prior to Vaccination 2 and to 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Initial Enrollment: Substudy B
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. When prevaccination assay results were lower than the LLOQ and the postvaccination results were greater than or equal to the LLOQ, the prevaccination assay results were set to LLOQ for the GMFR calculation.
Time Frame: From before vaccination 1 to prior to vaccination 2, 1, 4, and 8 weeks after the last vaccination (i.e., vaccination 1 and 2 for 1-visit schedule and 2 visit schedule, respectively)
Population: as for outcome 44
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
Fold Rise
  Prior to Vaccination 2: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A1 | 17.1 [6.1 to 48.1] | 6.5 [2.2 to 19.0] | 7.1 [2.6 to 19.1] | 6.0 [2.0 to 17.8] |  |  |  |  |  |  |
  Prior to Vaccination 2: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A2 | 5.7 [3.0 to 10.6] | 2.5 [1.3 to 4.8] | 2.9 [1.5 to 5.7] | 4.2 [2.0 to 8.9] |  |  |  |  |  |  |
  Prior to Vaccination 2: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B1 | 1.7 [1.1 to 2.7] | 2.0 [1.3 to 3.2] | 2.9 [1.4 to 6.2] | 3.2 [1.7 to 6.0] |  |  |  |  |  |  |
  Prior to Vaccination 2: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B2 | 1.4 [0.9 to 2.2] | 2.1 [1.1 to 4.1] | 2.1 [1.2 to 3.9] | 4.0 [1.8 to 9.1] |  |  |  |  |  |  |
  1 week after last vaccination: A1 | 24.8 [8.9 to 68.7] | 7.0 [2.8 to 17.6] | 10.3 [5.0 to 21.3] | 6.0 [2.2 to 16.3] | 6.0 [3.2 to 11.3] | 4.8 [1.8 to 13.3] | 3.6 [2.1 to 6.4] | 2.8 [1.3 to 6.0] | 3.6 [2.2 to 5.8] | 2.6 [1.6 to 4.3] | 2.8 [1.5 to 5.3]
  1 week after last vaccination: B1 | 2.3 [1.4 to 3.8] | 2.0 [1.4 to 2.8] | 2.6 [1.4 to 4.9] | 3.4 [2.0 to 5.6] | 2.0 [1.4 to 2.9] | 2.7 [1.6 to 4.5] | 1.2 [0.9 to 1.6] | 1.5 [1.0 to 2.3] | 1.6 [1.2 to 2.1] | 1.5 [1.2 to 1.8] | 1.8 [1.2 to 2.6]
  1 week after last vaccination: A2 | 6.5 [3.2 to 13.1] | 4.0 [2.5 to 6.4] | 4.0 [2.2 to 7.2] | 3.6 [1.8 to 7.2] | 1.7 [1.1 to 2.7] | 2.5 [1.0 to 6.4] | 2.3 [1.7 to 3.1] | 1.6 [0.9 to 2.7] | 4.8 [2.3 to 9.6] | 2.0 [1.3 to 3.1] | 2.4 [1.4 to 4.1]
  1 week after last vaccination: B2 | 1.6 [0.8 to 3.2] | 2.0 [1.1 to 3.7] | 2.1 [1.2 to 3.9] | 3.4 [1.7 to 6.6] | 1.9 [1.2 to 2.9] | 2.1 [2.1 to 3.3] | 1.2 [1.0 to 1.5] | 2.4 [1.2 to 4.9] | 1.2 [0.9 to 1.6] | 1.4 [1.0 to 1.9] | 1.4 [1.0 to 2.0]
  4 weeks after last vaccination: A1 | 14.6 [5.1 to 41.8] | 8.0 [3.0 to 21.6] | 10.3 [5.5 to 19.4] | 5.3 [2.0 to 14.0] | 8.0 [3.1 to 20.8] | 4.7 [1.8 to 12.6] | 10.1 [4.9 to 20.7] | 3.0 [1.5 to 5.9] | 5.2 [2.9 to 9.6] | 3.9 [2.2 to 7.1] | 6.6 [2.7 to 16.1]
  4 weeks after last vaccination: B1 | 3.2 [1.7 to 6.3] | 2.1 [1.6 to 2.8] | 2.3 [1.1 to 4.6] | 3.2 [1.7 to 6.0] | 3.2 [1.7 to 6.0] | 3.0 [1.5 to 6.0] | 2.5 [1.5 to 4.2] | 1.7 [1.2 to 2.5] | 1.7 [1.1 to 2.6] | 1.9 [1.4 to 2.7] | 2.2 [1.3 to 3.9]
  4 weeks after last vaccination: A2 | 3.5 [1.7 to 7.0] | 2.5 [1.8 to 3.4] | 3.5 [2.1 to 5.8] | 3.0 [1.8 to 5.0] | 3.8 [2.3 to 6.1] | 3.8 [2.3 to 6.3] | 4.4 [2.6 to 7.4] | 1.9 [1.2 to 3.1] | 5.0 [3.2 to 7.6] | 3.3 [2.1 to 5.2] | 7.6 [3.7 to 15.4]
  4 weeks after last vaccination: B2 | 1.7 [0.9 to 3.2] | 2.1 [1.2 to 3.7] | 1.5 [0.9 to 2.3] | 2.7 [1.4 to 5.2] | 2.7 [1.3 to 5.6] | 2.4 [1.3 to 4.4] | 1.8 [1.2 to 2.8] | 2.1 [1.0 to 4.5] | 1.2 [0.9 to 1.5] | 1.3 [0.9 to 1.8] | 1.5 [1.0 to 2.3]
  8 weeks after last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 15 | 12
  8 weeks after last vaccination: A1 | 13.0 [4.7 to 36.0] | 4.6 [2.0 to 10.6] | 5.5 [2.7 to 11.1] | 2.8 [1.1 to 7.3] | 6.0 [2.6 to 14.0] | 3.3 [1.1 to 10.4] | 6.6 [2.6 to 17.1] | 2.0 [1.1 to 3.7] | 5.8 [2.9 to 11.7] | 4.0 [2.0 to 8.1] | 6.0 [2.2 to 15.8]
  8 weeks after last vaccination: A2: number analyzed (Participants) | 10 | 10 | 10 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  8 weeks after last vaccination: A2 | 5.7 [2.8 to 11.5] | 3.7 [2.4 to 5.8] | 5.7 [3.3 to 9.7] | 3.0 [1.7 to 5.3] | 1.9 [1.1 to 3.3] | 2.1 [0.9 to 5.1] | 2.3 [1.1 to 4.9] | 0.6 [0.3 to 1.0] | 5.0 [2.4 to 10.3] | 3.1 [2.0 to 4.9] | 5.0 [2.7 to 9.5]
  8 weeks after last vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 15 | 12
  8 weeks after last vaccination: B1 | 2.5 [1.1 to 5.5] | 1.4 [0.9 to 2.2] | 1.9 [1.1 to 3.3] | 2.2 [1.3 to 3.8] | 2.5 [1.2 to 5.1] | 1.8 [0.7 to 4.2] | 1.0 [0.7 to 1.6] | 1.0 [0.6 to 1.5] | 1.6 [1.2 to 2.2] | 2.2 [1.5 to 3.4] | 2.4 [1.5 to 3.8]
  8 weeks after last vaccination: B2 | 1.3 [0.6 to 3.1] | 1.5 [0.8 to 3.0] | 1.6 [0.9 to 2.8] | 2.5 [1.3 to 4.9] | 2.1 [1.1 to 4.2] | 2.4 [1.1 to 5.3] | 1.7 [0.9 to 3.0] | 2.2 [1.2 to 4.1] | 1.2 [1.0 to 1.5] | 1.6 [1.1 to 2.3] | 1.4 [1.1 to 1.9]

48. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for Each Strain Prior to Vaccination 2 and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Expanded Enrollment: Substudy B
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Prior to vaccination 2 and at 1, 4, and 8 Weeks After last Vaccination
Population: EIP included all eligible participants who received vaccination; had blood drawn for assay testing within the specified time frame (26-35 days) after last vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. Here,'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Participants aged 65-85 years received a single intramuscular injection of qIRV dose level 1 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 98 | 108 | 105 | 24
Percentage of participants
  Prior to vaccination 2: A1: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to vaccination 2: A1 |  |  |  | 75.0 [53.3 to 90.2]
  Prior to vaccination 2: A2: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to vaccination 2: A2 |  |  |  | 79.2 [57.8 to 92.9]
  Prior to vaccination 2: B1: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to vaccination 2: B1 |  |  |  | 12.5 [2.7 to 32.4]
  Prior to vaccination 2: B2: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to vaccination 2: B2 |  |  |  | 8.3 [1.0 to 27.0]
  1 week after last vaccination: A1: number analyzed (Participants) | 96 | 106 | 105 | 24
  1 week after last vaccination: A1 | 40.6 [30.7 to 51.1] | 45.3 [35.6 to 55.2] | 39.0 [29.7 to 49.1] | 79.2 [57.8 to 92.9]
  1 week after last vaccination: B1: number analyzed (Participants) | 94 | 105 | 105 | 24
  1 week after last vaccination: B1 | 8.4 [3.7 to 15.9] | 12.1 [6.6 to 19.9] | 29.5 [21.0 to 39.2] | 79.2 [57.8 to 92.9]
  1 week after last vaccination: A2: number analyzed (Participants) | 96 | 107 | 105 | 24
  1 week after last vaccination: A2 | 22.3 [14.4 to 32.1] | 31.4 [22.7 to 41.2] | 21.9 [14.4 to 31.0] | 25.0 [9.8 to 46.7]
  1 week after last vaccination: B2: number analyzed (Participants) | 96 | 107 | 105 | 24
  1 week after last vaccination: B2 | 3.1 [0.6 to 8.9] | 7.5 [3.3 to 14.2] | 30.5 [21.9 to 40.2] | 16.7 [4.7 to 37.4]
  4 weeks after last vaccination: A1: number analyzed (Participants) | 98 | 107 | 105 | 24
  4 weeks after last vaccination: A1 | 55.1 [44.7 to 65.2] | 62.6 [52.7 to 71.8] | 49.5 [39.6 to 59.5] | 75.0 [53.3 to 90.2]
  4 weeks after last vaccination: B1: number analyzed (Participants) | 97 | 105 | 105 | 24
  4 weeks after last vaccination: B1 | 11.3 [5.8 to 19.4] | 20.4 [13.2 to 29.2] | 32.4 [23.6 to 42.2] | 87.5 [67.6 to 97.3]
  4 weeks after last vaccination: A2: number analyzed (Participants) | 97 | 108 | 105 | 24
  4 weeks after last vaccination: A2 | 40.2 [30.4 to 50.7] | 58.1 [48.1 to 67.7] | 29.5 [21.0 to 39.2] | 37.5 [18.8 to 59.4]
  4 weeks after last vaccination: B2: number analyzed (Participants) | 96 | 108 | 104 | 24
  4 weeks after last vaccination: B2 | 6.3 [2.3 to 13.1] | 12.0 [6.6 to 19.7] | 33.7 [24.7 to 43.6] | 16.7 [4.7 to 37.4]
  8 weeks after last vaccination: A1: number analyzed (Participants) | 98 | 106 | 105 | 24
  8 weeks after last vaccination: A1 | 59.2 [48.8 to 69.0] | 58.5 [48.5 to 68.0] | 37.1 [27.9 to 47.1] | 83.3 [62.6 to 95.3]
  8 weeks after last vaccination: A2: number analyzed (Participants) | 95 | 105 | 105 | 24
  8 weeks after last vaccination: A2 | 41.1 [31.1 to 51.6] | 50.5 [40.5 to 60.4] | 17.1 [10.5 to 25.7] | 75.0 [53.3 to 90.2]
  8 weeks after last vaccination: B1: number analyzed (Participants) | 97 | 107 | 105 | 24
  8 weeks after last vaccination: B1 | 4.1 [1.1 to 10.2] | 7.5 [3.3 to 14.2] | 18.1 [11.3 to 26.8] | 33.3 [15.6 to 55.3]
  8 weeks after last vaccination: B2: number analyzed (Participants) | 98 | 107 | 105 | 24
  8 weeks after last vaccination: B2 | 1.0 [0.0 to 5.6] | 1.9 [0.2 to 6.6] | 21.9 [14.4 to 31.0] | 12.5 [2.7 to 32.4]

49. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for Each Strain Prior to Vaccination 2 and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Initial Enrollment: Substudy B
Description: Seroconversion was defined as an HAI titer<1:10 prior to vaccination and>=1:40 at the time point of interest,or an HAI titer>=1:10 prior to vaccination with a 4-fold rise at the time point of interest.Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Prior to vaccination 2 (2-visit arms only), 1, 4 and 8 weeks after last vaccination (i.e., vaccination 1 for 1 visit and vaccination 2 for 2 visit)
Population: EIP=all eligible participants who received vaccination;had blood drawn for assay testing within specified time frame (26-35days)after Vaccination;had at least 1valid and determinate assay result at 4-week post-vaccination visit and had no major protocol deviations.All participants reported under'Overall Number of Participants Analyzed'contributed data to table;however,may not have evaluable data for every row and'Number Analyzed'signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 15 | 13 | 15 | 12
Percentage of participants
  Prior to Vaccination 2: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A1 | 90.0 [55.5 to 99.7] | 60.0 [26.2 to 87.8] | 63.6 [30.8 to 89.1] | 58.3 [27.7 to 84.8] |  |  |  |  |  |  |
  Prior to Vaccination 2: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A2 | 70.0 [34.8 to 93.3] | 50.0 [18.7 to 81.3] | 45.5 [16.7 to 76.6] | 50.0 [21.1 to 78.9] |  |  |  |  |  |  |
  Prior to Vaccination 2: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B1 | 10.0 [0.3 to 44.5] | 20.0 [2.5 to 55.6] | 45.5 [16.7 to 76.6] | 50.0 [21.1 to 78.9] |  |  |  |  |  |  |
  Prior to Vaccination 2: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B2 | 20.0 [2.5 to 55.6] | 30.0 [6.7 to 65.2] | 36.4 [10.9 to 69.2] | 50.0 [21.1 to 78.9] |  |  |  |  |  |  |
  1 week after last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  1 week after last vaccination: A1 | 90.0 [55.5 to 99.7] | 80.0 [44.4 to 97.5] | 90.9 [58.7 to 99.8] | 58.3 [27.7 to 84.8] | 75.0 [42.8 to 94.5] | 50.0 [21.1 to 78.9] | 66.7 [38.4 to 88.2] | 35.7 [12.8 to 64.9] | 58.3 [27.7 to 84.8] | 46.7 [21.3 to 73.4] | 50.0 [21.1 to 78.9]
  1 week after last vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  1 week after last vaccination: B1 | 40.0 [12.2 to 73.8] | 20.0 [2.5 to 55.6] | 45.5 [16.7 to 76.6] | 50.0 [21.1 to 78.9] | 33.3 [9.9 to 65.1] | 33.3 [9.9 to 65.1] | 6.7 [0.2 to 31.9] | 21.4 [4.7 to 50.8] | 7.7 [0.2 to 36.0] | 0.0 [0.0 to 23.2] | 25.0 [5.5 to 57.2]
  1 week after last vaccination: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  1 week after last vaccination: A2 | 80.0 [44.4 to 97.5] | 80.0 [44.4 to 97.5] | 63.6 [30.8 to 89.1] | 41.7 [15.2 to 72.3] | 16.7 [2.1 to 48.4] | 25.0 [5.5 to 57.2] | 26.7 [7.8 to 55.1] | 21.4 [4.7 to 50.8] | 66.7 [34.9 to 90.1] | 26.7 [7.8 to 55.1] | 33.3 [9.9 to 65.1]
  1 week after last vaccination: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  1 week after last vaccination: B2 | 20.0 [2.5 to 55.6] | 20.0 [2.5 to 55.6] | 36.4 [10.9 to 69.2] | 50.0 [21.1 to 78.9] | 25.0 [5.5 to 57.2] | 33.3 [9.9 to 65.1] | 0.0 [0.0 to 21.8] | 21.4 [4.7 to 50.8] | 7.7 [0.2 to 36.0] | 14.3 [1.8 to 42.8] | 16.7 [2.1 to 48.4]
  4 weeks after last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  4 weeks after last vaccination: A1 | 90.0 [55.5 to 99.7] | 80.0 [44.4 to 97.5] | 90.9 [58.7 to 99.8] | 41.7 [15.2 to 72.3] | 58.3 [27.7 to 84.8] | 50.0 [21.1 to 78.9] | 80.0 [51.9 to 95.7] | 35.7 [12.8 to 64.9] | 84.6 [54.6 to 98.1] | 60.0 [32.3 to 83.7] | 58.3 [27.7 to 84.8]
  4 weeks after vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  4 weeks after vaccination: B1 | 50.0 [18.7 to 81.3] | 20.0 [2.5 to 55.6] | 27.3 [6.0 to 61.0] | 50.0 [21.1 to 78.9] | 50.0 [21.1 to 78.9] | 41.7 [15.2 to 72.3] | 33.3 [11.8 to 61.6] | 14.3 [1.8 to 42.8] | 23.1 [5.0 to 53.8] | 28.6 [8.4 to 58.1] | 41.7 [15.2 to 72.3]
  4 weeks after last vaccination: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  4 weeks after last vaccination: A2 | 40.0 [12.2 to 73.8] | 20.0 [2.5 to 55.6] | 45.5 [16.7 to 76.6] | 50.0 [21.1 to 78.9] | 58.3 [27.7 to 84.8] | 58.3 [27.7 to 84.8] | 73.3 [44.9 to 92.2] | 28.6 [8.4 to 58.1] | 69.2 [38.6 to 90.9] | 53.3 [26.6 to 78.7] | 83.3 [51.6 to 97.9]
  4 weeks after last vaccination: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  4 weeks after last vaccination: B2 | 30.0 [6.7 to 65.2] | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 41.7 [15.2 to 72.3] | 25.0 [5.5 to 57.2] | 33.3 [9.9 to 65.1] | 20.0 [4.3 to 48.1] | 28.6 [8.4 to 58.1] | 7.7 [0.2 to 36.0] | 14.3 [1.8 to 42.8] | 25.0 [5.5 to 57.2]
  8 weeks after last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 15 | 12
  8 weeks after last vaccination: A1 | 80.0 [44.4 to 97.5] | 60.0 [26.2 to 87.8] | 72.7 [39.0 to 94.0] | 41.7 [15.2 to 72.3] | 58.3 [27.7 to 84.8] | 45.5 [16.7 to 76.6] | 73.3 [44.9 to 92.2] | 35.7 [12.8 to 64.9] | 84.6 [54.6 to 98.1] | 57.1 [28.9 to 82.3] | 63.6 [30.8 to 89.1]
  8 weeks after last vaccination: A2: number analyzed (Participants) | 10 | 10 | 10 | 12 | 11 | 11 | 15 | 14 | 13 | 14 | 12
  8 weeks after last vaccination: A2 | 70.0 [34.8 to 93.3] | 70.0 [34.8 to 93.3] | 80.0 [44.4 to 97.5] | 50.0 [21.1 to 78.9] | 9.1 [0.2 to 41.3] | 36.4 [10.9 to 69.2] | 46.7 [21.3 to 73.4] | 14.3 [1.8 to 42.8] | 69.2 [38.6 to 90.9] | 64.3 [35.1 to 87.2] | 83.3 [51.6 to 97.9]
  8 weeks after last vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 13 | 12
  8 weeks after last vaccination: B1 | 40.0 [12.2 to 73.8] | 10.0 [0.3 to 44.5] | 36.4 [10.9 to 69.2] | 33.3 [9.9 to 65.1] | 50.0 [21.1 to 78.9] | 36.4 [10.9 to 69.2] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 15.4 [1.9 to 45.4] | 38.5 [13.9 to 68.4] | 33.3 [9.9 to 65.1]
  8 weeks after last vaccination: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 13 | 12
  8 weeks after last vaccination: B2 | 20.0 [2.5 to 55.6] | 10.0 [0.3 to 44.5] | 9.1 [0.2 to 41.3] | 41.7 [15.2 to 72.3] | 25.0 [5.5 to 57.2] | 45.5 [16.7 to 76.6] | 20.0 [4.3 to 48.1] | 28.6 [8.4 to 58.1] | 0.0 [0.0 to 24.7] | 15.4 [1.9 to 45.4] | 8.3 [0.2 to 38.5]

50. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for Each Strain Before Vaccinations 1 and 2, and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Expanded Enrollment: Substudy B
Description: Proportion of participants achieving HAI titers >= 1:40 for each strain before vaccination and at 1, 4 and 8 weeks after vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination 1 and 2 and at 1, 4 and 8 weeks after last vaccination (i.e. after vaccination 1 for 1-vist schedule arms and after vaccination 2 for 2-visit schedule arms)
Population: EIP included all eligible participants who received vaccination;had blood drawn for assay testing within the specified time frame(26-35 days) after last vaccination;had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations.Here,Number Analyzed=participants evaluable for specified rows. All participants reported under 'Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, 65 to 85 Years: Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 2, dose combination 1 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-Visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 116 | 117 | 115 | 25
Percentage of participants
  Prior to vaccination 1: A1: number analyzed (Participants) | 98 | 107 | 105 | 24
  Prior to vaccination 1: A1 | 48.0 [37.8 to 58.3] | 51.4 [41.5 to 61.2] | 47.6 [37.8 to 57.6] | 33.3 [15.6 to 55.3]
  Prior to vaccination 1: A2: number analyzed (Participants) | 97 | 108 | 105 | 24
  Prior to vaccination 1: A2 | 67.0 [56.7 to 76.2] | 52.8 [42.9 to 62.5] | 54.3 [44.3 to 64.0] | 12.5 [2.7 to 32.4]
  Prior to vaccination 1: B1: number analyzed (Participants) | 97 | 108 | 105 | 24
  Prior to vaccination 1: B1 | 30.9 [21.9 to 41.1] | 33.3 [24.6 to 43.1] | 33.3 [24.4 to 43.2] | 8.3 [1.0 to 27.0]
  Prior to vaccination 1: B2: number analyzed (Participants) | 98 | 108 | 105 | 24
  Prior to vaccination 1: B2 | 23.5 [15.5 to 33.1] | 34.3 [25.4 to 44.0] | 23.8 [16.0 to 33.1] | 8.3 [1.0 to 27.0]
  Prior to vaccination 2: A1: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: A1 |  |  |  | 92.0 [74.0 to 99.0]
  Prior to vaccination 2: A2: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: A2 |  |  |  | 92.0 [74.0 to 99.0]
  Prior to vaccination 2: B1: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: B1 |  |  |  | 28.0 [12.1 to 49.4]
  Prior to vaccination 2: B2: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2: B2 |  |  |  | 20.0 [6.8 to 40.7]
  1 Week after last vaccination: A1: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 Week after last vaccination: A1 | 82.0 [73.1 to 89.0] | 84.1 [75.8 to 90.5] | 82.9 [74.3 to 89.5] | 96.0 [79.6 to 99.9]
  1 Week after last vaccination: B1: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 Week after last vaccination: B1 | 53.0 [42.8 to 63.1] | 54.2 [44.3 to 63.9] | 72.4 [62.8 to 80.7] | 44.0 [24.4 to 65.1]
  1 Week after last vaccination: A2: number analyzed (Participants) | 99 | 105 | 105 | 25
  1 Week after last vaccination: A2 | 86.9 [78.6 to 92.8] | 84.8 [76.4 to 91.0] | 84.8 [76.4 to 91.0] | 92.0 [74.0 to 99.0]
  1 Week after last vaccination: B2: number analyzed (Participants) | 100 | 107 | 105 | 25
  1 Week after last vaccination: B2 | 38.0 [28.5 to 48.3] | 40.2 [30.8 to 50.1] | 63.8 [53.9 to 73.0] | 28.0 [12.1 to 49.4]
  4 weeks after last vaccination: A1: number analyzed (Participants) | 105 | 110 | 108 | 25
  4 weeks after last vaccination: A1 | 88.6 [80.9 to 94.0] | 92.7 [86.2 to 96.8] | 86.1 [78.1 to 92.0] | 92.0 [74.0 to 99.0]
  4 weeks after last vaccination: B1: number analyzed (Participants) | 105 | 107 | 108 | 25
  4 weeks after last vaccination: B1 | 54.3 [44.3 to 64.0] | 60.9 [51.1 to 70.1] | 77.8 [68.8 to 85.2] | 52.0 [31.3 to 72.2]
  4 weeks after last vaccination: A2: number analyzed (Participants) | 105 | 110 | 108 | 25
  4 weeks after last vaccination: A2 | 94.3 [88.0 to 97.9] | 99.1 [94.9 to 100.0] | 88.9 [81.4 to 94.1] | 92.0 [74.0 to 99.0]
  4 weeks after last vaccination: B2: number analyzed (Participants) | 103 | 110 | 107 | 25
  4 weeks after last vaccination: B2 | 39.8 [30.3 to 49.9] | 50.0 [40.3 to 59.7] | 66.4 [56.6 to 75.2] | 28.0 [12.1 to 49.4]
  8 weeks after last vaccination: A1:: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after last vaccination: A1: | 89.5 [82.0 to 94.7] | 88.1 [80.5 to 93.5] | 75.0 [65.7 to 82.8] | 92.0 [74.0 to 99.0]
  8 weeks after last vaccination: A2:: number analyzed (Participants) | 103 | 107 | 108 | 25
  8 weeks after last vaccination: A2: | 94.2 [87.8 to 97.8] | 91.6 [84.6 to 96.1] | 58.3 [48.5 to 67.7] | 92.0 [74.0 to 99.0]
  8 weeks after last vaccination: B1:: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after last vaccination: B1: | 36.2 [27.0 to 46.1] | 41.3 [31.9 to 51.1] | 46.3 [36.7 to 56.2] | 44.0 [24.4 to 65.1]
  8 weeks after last vaccination: B2:: number analyzed (Participants) | 105 | 109 | 108 | 25
  8 weeks after last vaccination: B2: | 29.5 [21.0 to 39.2] | 29.4 [21.0 to 38.8] | 50.9 [41.1 to 60.7] | 24.0 [9.4 to 45.1]

51. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for Each Strain Before Vaccinations 1 and 2 and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Initial Enrollment: Substudy B
Description: Percentage of participants achieving HAI titers >= 1:40 for each strain before vaccinations 1 and 2 and at 1, 4 and 8 weeks after last vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination 1 and 2 (for 2-visit only), and 1, 4 and 8 weeks after last vaccination (i.e., vaccination 1 for 1-visit arms and vaccination 2 for 2-visit arms)
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in the opposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 15 | 13 | 15 | 12
Percentage of participants
  Prior to Vaccination 1: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  Prior to Vaccination 1: A1 | 40.0 [12.2 to 73.8] | 70.0 [34.8 to 93.3] | 63.6 [63.6 to 89.1] | 66.7 [34.9 to 90.1] | 50.0 [21.1 to 78.9] | 75.0 [42.8 to 94.5] | 53.3 [26.6 to 78.7] | 35.7 [12.8 to 64.9] | 69.2 [38.6 to 90.9] | 46.7 [21.3 to 73.4] | 66.7 [34.9 to 90.1]
  Prior to Vaccination 1: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  Prior to Vaccination 1: A2 | 70.0 [34.8 to 93.3] | 100.0 [69.2 to 100.0] | 72.7 [39.0 to 94.0] | 75.0 [42.8 to 94.5] | 83.3 [51.6 to 97.9] | 83.3 [51.6 to 97.9] | 66.7 [38.4 to 88.2] | 92.9 [66.1 to 99.8] | 30.8 [9.1 to 61.4] | 40.0 [16.3 to 67.7] | 50.0 [21.1 to 78.9]
  Prior to Vaccination 1: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  Prior to Vaccination 1: B1 | 30.0 [6.7 to 65.2] | 30.0 [6.7 to 65.2] | 45.5 [16.7 to 76.6] | 41.7 [15.2 to 72.3] | 33.3 [9.9 to 65.1] | 33.3 [9.9 to 65.1] | 13.3 [1.7 to 40.5] | 42.9 [17.7 to 71.1] | 15.4 [1.9 to 45.4] | 46.7 [21.3 to 73.4] | 25.0 [5.5 to 57.2]
  Prior to Vaccination 1: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  Prior to Vaccination 1: B2 | 10.0 [0.3 to 44.5] | 20.0 [2.5 to 55.6] | 18.2 [2.3 to 51.8] | 33.3 [9.9 to 65.1] | 25.0 [5.5 to 57.2] | 33.3 [9.9 to 65.1] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 23.1 [5.0 to 53.8] | 21.4 [4.7 to 50.8] | 33.3 [9.9 to 65.1]
  Prior to Vaccination 2: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A1 | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 90.9 [58.7 to 99.8] | 91.7 [61.5 to 99.8] |  |  |  |  |  |  |
  Prior to Vaccination 2: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: A2 | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7] | 90.9 [58.7 to 99.8] | 100.0 [73.5 to 100.0] |  |  |  |  |  |  |
  Prior to Vaccination 2: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B1 | 50.0 [18.7 to 81.3] | 60.0 [26.2 to 87.8] | 90.9 [58.7 to 99.8] | 91.7 [61.5 to 99.8] |  |  |  |  |  |  |
  Prior to Vaccination 2: B2: number analyzed (Participants) | 3 | 6 | 6 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2: B2 | 30.0 [6.7 to 65.2] | 60.0 [26.2 to 87.8] | 54.5 [23.4 to 83.3] | 83.3 [51.6 to 97.9] |  |  |  |  |  |  |
  1 week after the last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 12 | 15 | 12
  1 week after the last vaccination: A1 | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0] | 100.0 [73.5 to 100.0] | 100.0 [73.5 to 100.0] | 100.0 [73.5 to 100.0] | 93.3 [68.1 to 99.8] | 78.6 [49.2 to 95.3] | 83.3 [51.6 to 97.9] | 93.3 [68.1 to 99.8] | 91.7 [61.5 to 99.8]
  1 week after the last vaccination: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 12 | 15 | 12
  1 week after the last vaccination: A2 | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7] | 100.0 [71.5 to 100.0] | 91.7 [61.5 to 99.8] | 91.7 [61.5 to 99.8] | 100.0 [73.5 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [76.8 to 100.0] | 91.7 [61.5 to 99.8] | 80.0 [51.9 to 95.7] | 83.3 [51.6 to 97.9]
  1 week after the last vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  1 week after the last vaccination: B1 | 70.0 [34.8 to 93.3] | 80.0 [44.4 to 97.5] | 90.9 [58.7 to 99.8] | 91.7 [61.5 to 99.8] | 66.7 [34.9 to 90.1] | 83.3 [51.6 to 97.9] | 26.7 [7.8 to 55.1] | 64.3 [35.1 to 87.2] | 38.5 [13.9 to 68.4] | 60.0 [32.3 to 83.7] | 50.0 [21.1 to 78.9]
  1 week after the last vaccination: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  1 week after the last vaccination: B2 | 30.0 [6.7 to 65.2] | 60.0 [26.2 to 87.8] | 54.5 [23.4 to 83.3] | 83.3 [51.6 to 97.9] | 58.3 [27.7 to 84.8] | 66.7 [34.9 to 90.1] | 6.7 [0.2 to 31.9] | 21.4 [4.7 to 50.8] | 30.8 [9.1 to 61.4] | 33.3 [11.8 to 61.6] | 50.0 [21.1 to 78.9]
  4 weeks after the last vaccination: A1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 15 | 12
  4 weeks after the last vaccination: A1 | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0] | 91.7 [61.5 to 99.8] | 100.0 [73.5 to 100.0] | 100.0 [73.5 to 100.0] | 100.0 [78.2 to 100.0] | 85.7 [57.2 to 98.2] | 92.3 [64.0 to 99.8] | 93.3 [68.1 to 99.8] | 100.0 [73.5 to 100.0]
  4 weeks after the last vaccination: A2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 12 | 13 | 15 | 12
  4 weeks after the last vaccination: A2 | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0] | 100.0 [73.5 to 100.0] | 91.7 [61.5 to 99.8] | 100.0 [73.5 to 100.0] | 100.0 [78.2 to 100.0] | 85.7 [57.2 to 98.2] | 100.0 [75.3 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [73.5 to 100.0]
  4 weeks after the last vaccination: B1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  4 weeks after the last vaccination: B1 | 60.0 [26.2 to 87.8] | 70.0 [34.8 to 93.3] | 90.9 [58.7 to 99.8] | 83.3 [51.6 to 97.9] | 91.7 [61.5 to 99.8] | 75.0 [42.8 to 94.5] | 53.3 [26.6 to 78.7] | 71.4 [41.9 to 91.6] | 46.2 [19.2 to 74.9] | 78.6 [49.2 to 95.3] | 66.7 [34.9 to 90.1]
  4 weeks after the last vaccination: B2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  4 weeks after the last vaccination: B2 | 30.0 [6.7 to 65.2] | 40.0 [12.2 to 73.8] | 36.4 [10.9 to 69.2] | 66.7 [34.9 to 90.1] | 58.3 [27.7 to 84.8] | 58.3 [27.7 to 84.8] | 33.3 [11.8 to 61.6] | 35.7 [12.8 to 64.9] | 30.8 [9.1 to 61.4] | 42.9 [17.7 to 71.1] | 50.0 [21.1 to 78.9]
  8 weeks after the last vaccination: A1:: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 14 | 11
  8 weeks after the last vaccination: A1: | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 90.9 [58.7 to 99.8] | 83.3 [51.6 to 97.9] | 100.0 [73.5 to 100.0] | 100.0 [71.5 to 100.0] | 100.0 [78.2 to 100.0] | 64.3 [35.1 to 87.2] | 92.3 [64.0 to 99.8] | 92.9 [66.1 to 99.8] | 100.0 [71.5 to 100.0]
  8 weeks after the last vaccination: A2:: number analyzed (Participants) | 10 | 10 | 10 | 12 | 11 | 11 | 15 | 14 | 13 | 14 | 12
  8 weeks after the last vaccination: A2: | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 91.7 [61.5 to 99.8] | 90.9 [58.7 to 99.8] | 100.0 [71.5 to 100.0] | 93.3 [68.1 to 99.8] | 57.1 [28.9 to 82.3] | 92.3 [64.0 to 99.8] | 100.0 [76.8 to 100.0] | 100.0 [73.5 to 100.0]
  8 weeks after the last vaccination: B1:: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 14 | 12
  8 weeks after the last vaccination: B1: | 70.0 [34.8 to 93.3] | 50.0 [18.7 to 81.3] | 90.9 [58.7 to 99.8] | 75.0 [42.8 to 94.5] | 66.7 [34.9 to 90.1] | 45.5 [16.7 to 76.6] | 33.3 [11.8 to 61.6] | 35.7 [12.8 to 64.9] | 46.2 [19.2 to 74.9] | 78.6 [49.2 to 95.3] | 58.3 [27.7 to 84.8]
  8 weeks after the last vaccination: B2:: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 11 | 15 | 14 | 13 | 13 | 12
  8 weeks after the last vaccination: B2: | 30.0 [6.7 to 65.2] | 50.0 [18.7 to 81.3] | 27.3 [6.0 to 61.0] | 75.0 [42.8 to 94.5] | 50.0 [21.1 to 78.9] | 63.6 [30.8 to 89.1] | 33.3 [11.8 to 61.6] | 28.6 [8.4 to 58.1] | 30.8 [9.1 to 61.4] | 30.8 [9.1 to 61.4] | 58.3 [27.7 to 84.8]

52. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for All Strains Prior to Vaccination 2, and at 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Expanded Enrollment: Substudy B
Description: Seroconversion was defined as an HAI titer<1:10 prior to vaccination and>=1:40 at the time point of interest,or an HAI titer>=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Prior to vaccination 2 (for 2-visit schedule only) and at 1, 4, and 8 weeks after last vaccination (after vaccination 1 for 1-visit schedule and after vaccination 2 for 2-visit schedule)
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of qIRV dose level 1 as a part of expanded enrollment.
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 116 | 117 | 115 | 24
Percentage of participants
  Prior to vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 24
  Prior to vaccination 2 |  |  |  | 4.2 [0.1 to 21.1]
  1 week after last vaccination: number analyzed (Participants) | 93 | 104 | 105 | 24
  1 week after last vaccination | 0.0 [0.0 to 3.9] | 2.9 [0.6 to 8.2] | 10.5 [5.3 to 18.0] | 4.2 [0.1 to 21.1]
  4 weeks after last vaccination: number analyzed (Participants) | 94 | 104 | 104 | 24
  4 weeks after last vaccination | 3.2 [0.7 to 9.0] | 7.7 [3.4 to 14.6] | 13.5 [7.6 to 21.6] | 12.5 [2.7 to 32.4]
  8 weeks after last vaccination: number analyzed (Participants) | 95 | 104 | 105 | 24
  8 weeks after last vaccination | 1.1 [0.0 to 5.8] | 0.0 [0.0 to 3.5] | 4.8 [1.6 to 10.8] | 4.2 [0.1 to 21.1]

53. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for All Strains Prior to Vaccination 2 and at 1, 4, and 8 Weeks the Last Vaccination (Participants Aged 65-85 Years): Initial Enrollment: Substudy B
Description: as for outcome 52
Time Frame: as for outcome 52
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV followed by a single intramuscular injection of bIRV dose Level combination 1 administered 21 days apart as a part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 2-visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 15 | 13 | 14 | 12
Percentage of Participants
  Prior to Vaccination 2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prior to Vaccination 2 | 0.0 [0.0 to 3.8] | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 41.7 [15.2 to 72.3] |  |  |  |  |  |  |
  1 week after the last vaccination: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 11 | 14 | 12
  1 week after the last vaccination | 10.0 [0.3 to 44.5] | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 33.3 [9.9 to 65.1] | 0.0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 21.8] | 14.3 [1.8 to 42.8] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 23.2] | 16.7 [2.1 to 48.4]
  4 weeks after the last vaccination: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  4 weeks after the last vaccination | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8] | 9.1 [0.2 to 41.3] | 16.7 [2.1 to 48.4] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 20.0 [4.3 to 48.1] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 23.2] | 25.0 [5.5 to 57.2]
  8 weeks after the last vaccination: number analyzed (Participants) | 10 | 10 | 10 | 12 | 11 | 11 | 15 | 14 | 13 | 13 | 11
  8 weeks after the last vaccination | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8] | 25.0 [5.5 to 57.2] | 9.1 [0.2 to 41.3] | 18.2 [2.3 to 51.8] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 24.7] | 7.7 [0.2 to 36.0] | 9.1 [0.2 to 41.3]

54. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for All Strains Before Vaccinations 1 and 2 and 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Expanded Enrollment: Substudy B
Description: Percentage of participants with HAI titers >=1:40 for all strains before vaccinations 1 and 2 and 1, 4, and 8 weeks after the last vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Prior to vaccination 1 and 2, and at 1, 4, and 8 weeks after last vaccination (after vaccination 1 for 1-visit schedule and after vaccination 2 for 2-visit schedule)
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65-85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of Licensed QIV, 1-visit Schedule: Expanded Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Expanded Enrollment
Number analyzed (Participants) | 116 | 117 | 115 | 25
Percentage of participants
  Prior to vaccination 1: number analyzed (Participants) | 96 | 107 | 105 | 24
  Prior to vaccination 1 | 5.2 [1.7 to 11.7] | 12.1 [6.6 to 19.9] | 10.5 [5.3 to 18.0] | 0.0 [0.0 to 14.2]
  Prior to vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 25
  Prior to vaccination 2 |  |  |  | 12.0 [2.5 to 31.2]
  1 week after last vaccination: number analyzed (Participants) | 99 | 105 | 105 | 25
  1 week after last vaccination | 24.2 [16.2 to 33.9] | 26.7 [18.5 to 36.2] | 40.0 [30.6 to 50.0] | 16.0 [4.5 to 36.1]
  4 weeks after last vaccination: number analyzed (Participants) | 103 | 107 | 107 | 25
  4 weeks after last vaccination | 27.2 [18.9 to 36.8] | 36.4 [27.4 to 46.3] | 52.3 [42.5 to 62.1] | 20.0 [6.8 to 40.7]
  8 weeks after last vaccination: number analyzed (Participants) | 103 | 107 | 108 | 25
  8 weeks after last vaccination | 13.6 [7.6 to 21.8] | 13.1 [7.3 to 21.0] | 25.9 [18.0 to 35.2] | 12.0 [2.5 to 13.2]

55. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for All Strains Before Vaccinations 1 and 2 and 1, 4, and 8 Weeks After the Last Vaccination (Participants Aged 65-85 Years): Initial Enrollment: Substudy B
Description: as for outcome 54
Time Frame: Prior to vaccination 1 and 2 and at 1, 4, and 8 Weeks After the Last Vaccination (after vaccination 1 for 1-visit schedule and after vaccination 2 for 2-visit schedule)
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule 65-85 Years: Initial Enrollment: Participants aged 65 to 85 years received intramuscular injections with 2 doses qIRV at dose Level 1 administered 21 days apart as a part of initial enrollment.
- SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV administered concurrently in theopposite arm with a single intramuscular injection of bIRV AA (dose level combination 1) as part of initial enrollment.
Arm/Group | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule 65-85 Years: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment
Number analyzed (Participants) | 14 | 15 | 16 | 16 | 16 | 15 | 16 | 15 | 13 | 14 | 12
Percentage of participants
  Prior to Vaccination 1: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  Prior to Vaccination 1 | 10.0 [0.3 to 44.5] | 10.0 [0.3 to 44.5] | 18.2 [2.3 to 51.8] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4] | 6.7 [0.2 to 31.9] | 7.1 [0.2 to 33.9] | 7.7 [0.2 to 36.0] | 7.1 [0.2 to 33.9] | 25.0 [5.5 to 57.2]
  Prior to Vaccination 2: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  Prior to Vaccination 2 | 30.0 [6.7 to 65.2] | 50.0 [18.7 to 81.3] | 54.5 [23.4 to 83.3] | 66.7 [34.9 to 90.1] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  1 Week after the last vaccination: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  1 Week after the last vaccination | 20.0 [2.5 to 55.6] | 60.0 [26.2 to 87.8] | 54.5 [23.4 to 83.3] | 66.7 [34.9 to 90.1] | 41.7 [15.2 to 72.3] | 58.3 [27.7 to 84.8] | 6.7 [0.2 to 31.9] | 14.3 [1.8 to 42.8] | 27.3 [6.0 to 61.0] | 13.3 [1.7 to 40.5] | 41.7 [15.2 to 72.3]
  4 Weeks after the last vaccination: number analyzed (Participants) | 10 | 10 | 11 | 12 | 12 | 12 | 15 | 14 | 13 | 14 | 12
  4 Weeks after the last vaccination | 20.0 [2.5 to 55.6] | 40.0 [12.2 to 73.8] | 36.4 [10.9 to 69.2] | 66.7 [34.9 to 90.1] | 50.0 [21.1 to 78.9] | 58.3 [27.7 to 84.8] | 33.3 [11.8 to 61.6] | 21.4 [4.7 to 50.8] | 23.1 [5.0 to 53.8] | 35.7 [12.8 to 64.9] | 41.7 [15.2 to 72.3]
  8 Weeks after the last vaccination: number analyzed (Participants) | 10 | 10 | 10 | 12 | 11 | 11 | 15 | 14 | 13 | 14 | 12
  8 Weeks after the last vaccination | 20.0 [2.5 to 55.6] | 40.0 [12.2 to 73.8] | 20.0 [2.5 to 55.6] | 50.0 [21.1 to 78.9] | 45.5 [16.7 to 76.6] | 45.5 [16.7 to 76.6] | 20.0 [4.3 to 48.1] | 7.1 [0.2 to 33.9] | 15.4 [1.9 to 45.4] | 30.8 [9.1 to 61.4] | 45.5 [16.7 to 76.6]

56. Secondary Outcome: HAI GMTs Before Vaccination and at 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: HAI GMT before vaccination and at 1, 4, and 8 weeks after vaccination was described in this outcome measure. GMTs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution).
Time Frame: Before vaccination and 1, 4, and 8 Weeks After the Vaccination
Population: as for outcome 49
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 128 | 129
Titers
  Prior to vaccination: A1: number analyzed (Participants) | 112 | 110
  Prior to vaccination: A1 | 21.4 [16.8 to 27.3] | 18.0 [14.4 to 22.5]
  Prior to vaccination: A2: number analyzed (Participants) | 112 | 110
  Prior to vaccination: A2 | 16.5 [13.4 to 20.4] | 13.2 [11.0 to 15.8]
  Prior to vaccination: B1: number analyzed (Participants) | 112 | 109
  Prior to vaccination: B1 | 22.1 [17.7 to 27.6] | 19.0 [15.7 to 23.0]
  Prior to vaccination: B2: number analyzed (Participants) | 112 | 110
  Prior to vaccination: B2 | 11.6 [9.7 to 13.8] | 11.6 [9.8 to 13.6]
  1 week after vaccination: A1: number analyzed (Participants) | 113 | 110
  1 week after vaccination: A1 | 113.0 [85.3 to 149.7] | 124.6 [95.2 to 163.2]
  1 week after vaccination: A2: number analyzed (Participants) | 113 | 110
  1 week after vaccination: A2 | 52.7 [41.4 to 67.1] | 72.3 [57.3 to 91.3]
  1 week after vaccination: B1: number analyzed (Participants) | 112 | 110
  1 week after vaccination: B1 | 39.3 [31.3 to 49.2] | 37.1 [29.8 to 46.2]
  1 week after vaccination: B2: number analyzed (Participants) | 112 | 110
  1 week after vaccination: B2 | 16.0 [13.3 to 19.2] | 19.0 [15.7 to 23.1]
  4 weeks after vaccination: A1: number analyzed (Participants) | 113 | 108
  4 weeks after vaccination: A1 | 317.3 [251.8 to 399.8] | 273.6 [215.9 to 346.8]
  4 weeks after vaccination: A2: number analyzed (Participants) | 113 | 109
  4 weeks after vaccination: A2 | 140.9 [118.1 to 168.2] | 148.2 [123.9 to 177.4]
  4 weeks after vaccination: B1: number analyzed (Participants) | 113 | 108
  4 weeks after vaccination: B1 | 58.9 [48.8 to 71.1] | 48.2 [39.6 to 58.7]
  4 weeks after vaccination: B2: number analyzed (Participants) | 112 | 110
  4 weeks after vaccination: B2 | 19.8 [16.4 to 23.8] | 23.3 [19.1 to 28.3]
  8 weeks after vaccination: A1: number analyzed (Participants) | 111 | 109
  8 weeks after vaccination: A1 | 228.9 [183.2 to 285.9] | 221.2 [176.2 to 277.8]
  8 weeks after vaccination: A2: number analyzed (Participants) | 105 | 109
  8 weeks after vaccination: A2 | 80.0 [64.3 to 99.5] | 92.6 [76.4 to 112.2]
  8 weeks after vaccination: B1: number analyzed (Participants) | 111 | 109
  8 weeks after vaccination: B1 | 39.0 [32.0 to 47.6] | 34.8 [27.8 to 43.5]
  8 weeks after vaccination: B2: number analyzed (Participants) | 110 | 107
  8 weeks after vaccination: B2 | 17.9 [14.8 to 21.5] | 19.1 [15.8 to 23.2]

57. Secondary Outcome: HAI GMFR From Before Vaccination to 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. When prevaccination assay results were lower than the LLOQ and the postvaccination results were greater than or equal to the LLOQ, the pre vaccination assay results were set to LLOQ for the GMFR calculation.
Time Frame: Before vaccination to 1, 4, and 8 Weeks After Vaccination
Population: as for outcome 49
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 113 | 110
Fold Rise
  1 Week after vaccination: A1: number analyzed (Participants) | 112 | 110
  1 Week after vaccination: A1 | 4.5 [3.6 to 5.6] | 5.7 [4.5 to 7.2]
  1 Week after vaccination: A2: number analyzed (Participants) | 112 | 110
  1 Week after vaccination: A2 | 2.7 [2.3 to 3.3] | 4.4 [3.6 to 5.4]
  1 Week after vaccination: B1: number analyzed (Participants) | 111 | 109
  1 Week after vaccination: B1 | 1.7 [1.5 to 1.9] | 1.8 [1.6 to 2.1]
  1 Week after vaccination: B2: number analyzed (Participants) | 111 | 110
  1 Week after vaccination: B2 | 1.2 [1.1 to 1.3] | 1.4 [1.3 to 1.6]
  4 Weeks after vaccination: A1: number analyzed (Participants) | 112 | 108
  4 Weeks after vaccination: A1 | 12.3 [9.6 to 15.7] | 12.2 [9.5 to 15.6]
  4 Weeks after vaccination: A2: number analyzed (Participants) | 112 | 109
  4 Weeks after vaccination: A2 | 6.8 [5.7 to 8.2] | 8.7 [7.1 to 10.6]
  4 Weeks after vaccination: B1: number analyzed (Participants) | 112 | 108
  4 Weeks after vaccination: B1 | 2.4 [2.1 to 2.8] | 2.2 [1.9 to 2.6]
  4 Weeks after vaccination: B2: number analyzed (Participants) | 111 | 110
  4 Weeks after vaccination: B2 | 1.4 [1.3 to 1.6] | 1.7 [1.5 to 2.0]
  8 Weeks after vaccination: A1: number analyzed (Participants) | 110 | 109
  8 Weeks after vaccination: A1 | 8.9 [7.1 to 11.3] | 9.9 [8.0 to 12.4]
  8 Weeks after vaccination: A2: number analyzed (Participants) | 104 | 109
  8 Weeks after vaccination: A2 | 3.9 [3.2 to 4.9] | 5.5 [4.6 to 6.5]
  8 Weeks after vaccination: B1: number analyzed (Participants) | 110 | 108
  8 Weeks after vaccination: B1 | 1.7 [1.5 to 1.9] | 1.7 [1.4 to 1.9]
  8 Weeks after vaccination: B2: number analyzed (Participants) | 109 | 107
  8 Weeks after vaccination: B2 | 1.3 [1.2 to 1.4] | 1.4 [1.3 to 1.6]

58. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for Each Strain at 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: as for outcome 52
Time Frame: 1, 4, and 8 Weeks After Vaccination
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 131 | 131
Percentage of participants
  1 Week after vaccination: A1: number analyzed (Participants) | 112 | 110
  1 Week after vaccination: A1 | 57.1 [47.4 to 66.5] | 65.5 [55.8 to 74.3]
  1 Week after vaccination: A2: number analyzed (Participants) | 112 | 110
  1 Week after vaccination: A2 | 51.8 [42.1 to 61.3] | 58.2 [48.4 to 67.5]
  1 Week after vaccination: B1: number analyzed (Participants) | 111 | 109
  1 Week after vaccination: B1 | 23.4 [15.9 to 32.4] | 26.6 [18.6 to 35.9]
  1 Week after vaccination: B2: number analyzed (Participants) | 111 | 110
  1 Week after vaccination: B2 | 5.4 [2.0 to 11.4] | 12.7 [7.1 to 20.4]
  4 Weeks after vaccination: A1: number analyzed (Participants) | 112 | 108
  4 Weeks after vaccination: A1 | 83.0 [74.8 to 89.5] | 88.9 [81.4 to 94.1]
  4 Weeks after vaccination: A2: number analyzed (Participants) | 112 | 109
  4 Weeks after vaccination: A2 | 80.4 [71.8 to 87.3] | 89.0 [81.6 to 94.2]
  4 Weeks after vaccination: B1: number analyzed (Participants) | 112 | 108
  4 Weeks after vaccination: B1 | 40.2 [31.0 to 49.9] | 32.4 [23.7 to 42.1]
  4 Weeks after vaccination: B2: number analyzed (Participants) | 112 | 110
  4 Weeks after vaccination: B2 | 11.7 [6.4 to 19.2] | 21.8 [14.5 to 30.7]
  8 Weeks after vaccination: A1: number analyzed (Participants) | 110 | 109
  8 Weeks after vaccination: A1 | 79.1 [70.3 to 86.3] | 86.2 [78.3 to 92.1]
  8 Weeks after vaccination: A2: number analyzed (Participants) | 104 | 109
  8 Weeks after vaccination: A2 | 60.6 [50.5 to 70.0] | 76.1 [67.0 to 83.8]
  8 Weeks after vaccination: B1: number analyzed (Participants) | 110 | 108
  8 Weeks after vaccination: B1 | 22.7 [15.3 to 31.7] | 21.3 [14.0 to 30.2]
  8 Weeks after vaccination: B2: number analyzed (Participants) | 109 | 107
  8 Weeks after vaccination: B2 | 9.2 [4.5 to 16.2] | 10.3 [5.2 to 17.7]

59. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for Each Strain Before Vaccination and at 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: Percentage of participants with HAI titers >=1:40 for each strain before vaccination and 1, 4, and 8 weeks after vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination and 1, 4, and 8 Weeks After Vaccination
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 131 | 131
Percentage of participants
  Prior to vaccination: A1: number analyzed (Participants) | 112 | 110
  Prior to vaccination: A1 | 39.3 [30.2 to 49.0] | 35.5 [26.6 to 45.1]
  Prior to vaccination: A2: number analyzed (Participants) | 112 | 110
  Prior to vaccination: A2 | 34.8 [26.1 to 44.4] | 24.5 [16.8 to 33.7]
  Prior to vaccination: B1: number analyzed (Participants) | 112 | 109
  Prior to vaccination: B1 | 35.7 [26.9 to 45.3] | 37.6 [28.5 to 47.4]
  Prior to vaccination: B2: number analyzed (Participants) | 112 | 110
  Prior to vaccination: B2 | 17.9 [11.3 to 26.2] | 17.3 [10.7 to 25.7]
  1 Week after vaccination: A1: number analyzed (Participants) | 113 | 110
  1 Week after vaccination: A1 | 82.3 [74.0 to 88.8] | 81.8 [73.3 to 88.5]
  1 Week after vaccination: A2: number analyzed (Participants) | 113 | 110
  1 Week after vaccination: A2 | 75.2 [66.2 to 82.9] | 79.1 [70.3 to 86.3]
  1 Week after vaccination: B1: number analyzed (Participants) | 112 | 110
  1 Week after vaccination: B1 | 61.6 [51.9 to 70.6] | 53.6 [43.9 to 63.2]
  1 Week after vaccination: B2: number analyzed (Participants) | 29 | 39
  1 Week after vaccination: B2 | 25.9 [18.1 to 35.0] | 35.5 [26.6 to 45.1]
  4 Weeks after vaccination: A1: number analyzed (Participants) | 112 | 110
  4 Weeks after vaccination: A1 | 94.7 [88.8 to 98.0] | 96.3 [90.8 to 99.0]
  4 Weeks after vaccination: A2: number analyzed (Participants) | 113 | 109
  4 Weeks after vaccination: A2 | 98.2 [93.8 to 99.8] | 95.4 [89.6 to 98.5]
  4 Weeks after vaccination: B1: number analyzed (Participants) | 113 | 108
  4 Weeks after vaccination: B1 | 77.9 [69.1 to 85.1] | 63.9 [54.1 to 72.9]
  4 Weeks after vaccination: B2: number analyzed (Participants) | 112 | 110
  4 Weeks after vaccination: B2 | 33.9 [25.3 to 43.5] | 47.3 [37.7 to 57.0]
  8 Weeks after vaccination: A1: number analyzed (Participants) | 111 | 109
  8 Weeks after vaccination: A1 | 94.6 [88.6 to 98.0] | 95.4 [89.6 to 98.5]
  8 Weeks after vaccination: A2: number analyzed (Participants) | 105 | 109
  8 Weeks after vaccination: A2 | 86.7 [78.6 to 92.5] | 90.8 [83.8 to 95.5]
  8 Weeks after vaccination: B1: number analyzed (Participants) | 111 | 109
  8 Weeks after vaccination: B1 | 61.3 [51.5 to 70.4] | 53.2 [43.4 to 62.8]
  8 Weeks after vaccination: B2: number analyzed (Participants) | 110 | 107
  8 Weeks after vaccination: B2 | 28.2 [20.0 to 37.6] | 37.4 [28.2 to 47.3]

60. Secondary Outcome: Percentage of Participants Achieving HAI Seroconversion for All Strains at 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: as for outcome 52
Time Frame: 1, 4, and 8 Weeks After Vaccination
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 131 | 131
Percentage of participants
  1 Week after vaccination: number analyzed (Participants) | 110 | 109
  1 Week after vaccination | 1.8 [0.2 to 6.4] | 4.6 [1.5 to 10.4]
  4 Weeks after vaccination: number analyzed (Participants) | 111 | 107
  4 Weeks after vaccination | 7.2 [3.2 to 13.7] | 9.3 [4.6 to 16.5]
  8 Weeks after vaccination: number analyzed (Participants) | 103 | 106
  8 Weeks after vaccination | 3.9 [1.1 to 9.6] | 4.7 [1.5 to 10.7]

61. Secondary Outcome: Percentage of Participants With HAI Titers >=1:40 for All Strains Before Vaccination and 1, 4, and 8 Weeks After Vaccination (Participants Aged 18-64 Years): Substudy B
Description: Percentage of participants with HAI titers >=1:40 for all strains before vaccination and 1, 4, and 8 weeks after vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method.
Time Frame: Before vaccination and 1, 4, and 8 Weeks After Vaccination
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years: Expanded Enrollment
Number analyzed (Participants) | 131 | 131
Percentage of participants
  Prior to vaccination: number analyzed (Participants) | 112 | 109
  Prior to vaccination | 6.3 [2.5 to 12.5] | 1.8 [0.2 to 6.5]
  1 Week after vaccination: number analyzed (Participants) | 111 | 110
  1 Week after vaccination | 15.3 [9.2 to 23.4] | 20.9 [13.7 to 29.7]
  4 Weeks after vaccination: number analyzed (Participants) | 112 | 107
  4 Weeks after vaccination | 26.8 [18.9 to 36.0] | 32.7 [24.0 to 42.5]
  8 Weeks after vaccination: number analyzed (Participants) | 104 | 107
  8 Weeks after vaccination | 14.4 [8.3 to 22.7] | 22.4 [14.9 to 31.5]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events(Systematic assessment): from Day 1 to Day 7 after vaccination 1 and/or 2;Non-systematic assessment: SAEs: from vaccination 1 up to 6 months after last vaccination: other AEs: from vaccination 1 up to 4 weeks after last vaccination (After vaccination 2 for SSA arms and SSB 2-visit schedule arms and after vaccination 1 for SSB 1-visit schedule arms).
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both AE and non-SAE.
Groups:
- SSB: 1 Dose of QIV, 1 Visit Schedule, Expanded Enrollment: Participants aged 65 to 85 years received a single intramuscular injection of licensed QIV as a part of expanded enrollment.
- SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule, Expanded Enrollment: Participants aged 65 to 85 years received intramuscular injections with 2 doses qIRV at dose Level 1 administered 21 days apart as a part of expanded enrollment.
Arm/Group | SSA: mIRV A (Dose Level 1) + QIV | SSA: mIRV A (Dose Level 2) + QIV | SSA: mIRV A (Dose Level 3) + QIV | SSA: mIRV A (Dose Level 4) + QIV | SSA: mIRV A - Licensed QIV | SSA: mIRV B (Dose Level 1) + QIV | SSA: mIRV B (Dose Level 2) + QIV | SSA: mIRV B (Dose Level 3) + QIV | SSA: mIRV B (Dose Level 4) + QIV | SSA: mIRV B - Licensed QIV | SSA: bIRV AB (Dose Level Combination 1) + QIV | SSA: bIRV AB (Dose Level Combination 2) + QIV | SSA: bIRV AB (Dose Level Combination 3) + QIV | SSA: bIRV AB (Dose Level Combination 4) + QIV | SSA: bIRV AB-Licensed QIV | SSA: qIRV (Dose Level 1) + QIV | SSA: qIRV - Licensed QIV | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment | SSB: 1 Dose of QIV, 1 Visit Schedule, Expanded Enrollment | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule, Expanded Enrollment
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/14 | 0/15 | 0/17 | 0/14 | 0/15 | 0/14 | 0/15 | 0/14 | 0/16 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 0/16 | 0/16 | 0/16 | 0/15 | 0/16 | 0/15 | 0/131 | 0/131 | 0/116 | 0/117 | 0/115 | 0/14 | 0/16 | 0/15 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/14 | 0/15 | 1/17 | 0/14 | 0/15 | 0/14 | 1/15 | 1/14 | 0/16 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14 | 0/15 | 0/16 | 0/16 | 1/16 | 0/15 | 0/16 | 0/15 | 0/131 | 2/131 | 1/116 | 0/117 | 0/115 | 0/14 | 0/16 | 0/15 | 0/117
Other Adverse Events (participants affected / at risk) | 9/16 | 9/15 | 7/14 | 9/14 | 11/15 | 9/17 | 8/14 | 9/15 | 8/14 | 12/15 | 9/14 | 9/16 | 11/15 | 11/15 | 11/15 | 13/15 | 12/15 | 12/14 | 11/15 | 9/16 | 9/16 | 10/16 | 10/15 | 8/16 | 7/15 | 87/131 | 92/131 | 71/116 | 76/117 | 52/115 | 6/14 | 7/16 | 8/15 | 82/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SSA: mIRV A (Dose Level 1) + QIV (N=16) | SSA: mIRV A (Dose Level 2) + QIV (N=15) | SSA: mIRV A (Dose Level 3) + QIV (N=14) | SSA: mIRV A (Dose Level 4) + QIV (N=14) | SSA: mIRV A - Licensed QIV (N=15) | SSA: mIRV B (Dose Level 1) + QIV (N=17) | SSA: mIRV B (Dose Level 2) + QIV (N=14) | SSA: mIRV B (Dose Level 3) + QIV (N=15) | SSA: mIRV B (Dose Level 4) + QIV (N=14) | SSA: mIRV B - Licensed QIV (N=15) | SSA: bIRV AB (Dose Level Combination 1) + QIV (N=14) | SSA: bIRV AB (Dose Level Combination 2) + QIV (N=16) | SSA: bIRV AB (Dose Level Combination 3) + QIV (N=15) | SSA: bIRV AB (Dose Level Combination 4) + QIV (N=15) | SSA: bIRV AB-Licensed QIV (N=15) | SSA: qIRV (Dose Level 1) + QIV (N=15) | SSA: qIRV - Licensed QIV (N=15) | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment (N=14) | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment (N=15) | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment (N=16) | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment (N=16) | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment (N=16) | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment (N=15) | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment (N=16) | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment (N=15) | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment (N=131) | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment (N=131) | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment (N=116) | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment (N=117) | SSB: 1 Dose of QIV, 1 Visit Schedule, Expanded Enrollment (N=115) | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment (N=14) | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment (N=16) | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment (N=15) | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule, Expanded Enrollment (N=117)
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SSA: mIRV A (Dose Level 1) + QIV (N=16) | SSA: mIRV A (Dose Level 2) + QIV (N=15) | SSA: mIRV A (Dose Level 3) + QIV (N=14) | SSA: mIRV A (Dose Level 4) + QIV (N=14) | SSA: mIRV A - Licensed QIV (N=15) | SSA: mIRV B (Dose Level 1) + QIV (N=17) | SSA: mIRV B (Dose Level 2) + QIV (N=14) | SSA: mIRV B (Dose Level 3) + QIV (N=15) | SSA: mIRV B (Dose Level 4) + QIV (N=14) | SSA: mIRV B - Licensed QIV (N=15) | SSA: bIRV AB (Dose Level Combination 1) + QIV (N=14) | SSA: bIRV AB (Dose Level Combination 2) + QIV (N=16) | SSA: bIRV AB (Dose Level Combination 3) + QIV (N=15) | SSA: bIRV AB (Dose Level Combination 4) + QIV (N=15) | SSA: bIRV AB-Licensed QIV (N=15) | SSA: qIRV (Dose Level 1) + QIV (N=15) | SSA: qIRV - Licensed QIV (N=15) | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule: Initial Enrollment (N=14) | SSB: Licensed QIV + bIRV AA (Dose Level Combination 1), 2- Visit Schedule: Initial Enrollment (N=15) | SSB: Licensed QIV + bIRV AA (Dose Level Combination 2), 2- Visit Schedule: Initial Enrollment (N=16) | SSB: 2 Doses of Licensed QIV, 2-visit Schedule: Initial Enrollment (N=16) | SSB: Licensed QIV +bIRV AA (Dose Level Combination 1), 1-visit Schedule: Initial Enrollment (N=16) | SSB: Licensed QIV +bIRV AA (Dose Level Combination 2), 1-visit Schedule: Initial Enrollment (N=15) | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule: Initial Enrollment (N=16) | SSB: 1 Dose of Licensed QIV, 1 Visit Schedule: Initial Enrollment (N=15) | SSB: qIRV (Dose Level 1), 1-visit Schedule, 18-64 Years: Expanded Enrollment (N=131) | SSB: qIRV (Dose Level 2), 1-visit Schedule, 18-64 Years : Expanded Enrollment (N=131) | SSB: qIRV (Dose Level 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment (N=116) | SSB: qIRV (Dose Level 2, Dose Combination 1), 1-visit Schedule, 65 to 85 Years: Expanded Enrollment (N=117) | SSB: 1 Dose of QIV, 1 Visit Schedule, Expanded Enrollment (N=115) | SSB: bIRV AA + bIRV BB ( Both Dose Level Combination 1), 1-visit Schedule: Initial Enrollment (N=14) | SSB: qIRV (Dose Level 2, Dose Combination 2), 1-Visit Schedule: Initial Enrollment (N=16) | SSB: qIRV (Dose Level 3), 1-Visit Schedule: Initial Enrollment (N=15) | SSB: 2 Doses qIRV (Dose Level 1), 2 Visit Schedule, Expanded Enrollment (N=117)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 9 | 5 | 5 | 6 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (REDNESS) (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 13 | 16 | 4 | 9 | 5 | 2 | 1 | 4 | 14
Injection site pain (PAIN) (General disorders) | 4 | 5 | 7 | 9 | 8 | 6 | 4 | 7 | 5 | 7 | 6 | 5 | 9 | 7 | 6 | 13 | 10 | 8 | 8 | 6 | 6 | 6 | 9 | 8 | 2 | 79 | 82 | 51 | 68 | 32 | 4 | 6 | 6 | 68
Injection site swelling (SWELLING) (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 13 | 22 | 12 | 12 | 6 | 2 | 3 | 1 | 18
Pyrexia (FEVER) (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5 | 11 | 4 | 7 | 3 | 1 | 1 | 2 | 6
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 1 | 4 | 1 | 2 | 1 | 1 | 3 | 2 | 2 | 3 | 1 | 2 | 1 | 1 | 24 | 23 | 15 | 20 | 1 | 3 | 0 | 3 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 2 | 2 | 1 | 3 | 2 | 3 | 4 | 2 | 3 | 5 | 2 | 2 | 3 | 3 | 4 | 5 | 2 | 5 | 5 | 4 | 2 | 5 | 3 | 4 | 3 | 50 | 47 | 24 | 32 | 12 | 3 | 1 | 3 | 31
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 6 | 2 | 1 | 1 | 8
Chills (CHILLS) (General disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 1 | 4 | 0 | 1 | 2 | 1 | 5 | 5 | 2 | 0 | 2 | 2 | 2 | 1 | 25 | 27 | 8 | 21 | 5 | 2 | 0 | 2 | 23
Fatigue (FATIGUE) (General disorders) | 5 | 2 | 2 | 5 | 1 | 3 | 2 | 3 | 5 | 6 | 5 | 4 | 6 | 7 | 4 | 6 | 8 | 7 | 7 | 4 | 5 | 5 | 5 | 4 | 5 | 57 | 54 | 38 | 49 | 24 | 3 | 4 | 4 | 42
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 5 | 1 | 1 | 1 | 2 | 4 | 2 | 1 | 2 | 4 | 3 | 5 | 1 | 36 | 42 | 19 | 25 | 9 | 3 | 1 | 3 | 25
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (3):
  • Study Protocol (2022-07-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT05052697/Prot_000.pdf
  • Statistical Analysis Plan: Sub Study A (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT05052697/SAP_001.pdf
  • Statistical Analysis Plan: Sub Study B (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT05052697/SAP_002.pdf